CLINICAL TRIAL: NCT02407236
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Protocol to Evaluate the Safety and Efficacy of Ustekinumab Induction and Maintenance Therapy in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study to Evaluate the Safety and Efficacy of Ustekinumab Induction and Maintenance Therapy in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: UNIFI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CR106920; 2014-005606-38 (EudraCT Number); CNTO1275UCO3001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Results first posted 2019-12-23 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Colitis, Ulcerative; Inflammatory Bowel Diseases
Keywords: Ustekinumab; Inflammatory Bowel Diseases (IBD); Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (10):
- Induction Study - Placebo Intravenous (IV) (Placebo Comparator): Participants will be randomized to receive single dose of placebo as Intravenous (IV: into the vein) infusion at Week 0. Participants with clinical response at Week 8 will be eligible to enter the Maintenance study, but will not be randomized.
  Interventions: Drug: Placebo IV
- Induction Study - Ustekinumab 130 milligram (mg) IV (Experimental): Participants will be randomized to receive single dose of ustekinumab 130 mg as IV infusion at Week 0. Participants with clinical response at Week 8 will be eligible to enter the Maintenance study and will be randomized.
  Interventions: Drug: Ustekinumab IV
- Induction Study - Ustekinumab 6 mg/kg IV (Experimental): Participants will be randomized to receive ustekinumab approximating 6 mg/kg of body weight, as intravenous infusion at Week 0. Participants with clinical response at Week 8 will be eligible to enter the Maintenance study and will be randomized.
  Interventions: Drug: Ustekinumab IV
- Induction Study- Placebo- Nonresponsders at Week 8 (Other): Participants without clinical response to placebo at Week 8 will receive a single IV infusion of ustekinumab approximating 6mg/kg along with matching subcutaneous (SC) placebo (to maintain the blind). Participants in clinical response at Week 16 will be eligible to enter Maintenance study and will be randomized.
  Interventions: Drug: Placebo SC; Drug: Ustekinumab IV
- Induction study-Ustekinumab Nonresponders at Week 8 (Other): Participants without clinical response to ustekinumab (130 mg or 6 mg/kg [IV]) at Week 8 will receive a single dose of ustekinumab 90 mg subcutaneously along with matching placebo intravenously (to maintain the blind). Participants in clinical response at Week 16 (that is, delayed responders) will be eligible to enter Maintenance study, but will not be randomized.
  Interventions: Drug: Placebo IV; Drug: Ustekinumab SC
- Maintenance Study - Placebo Subcutaneous (SC) (Placebo Comparator): Participants in clinical response (at Week 8 or Week 16) to Induction treatment with single IV infusion of Ustekinumab will be randomized to receive placebo subcutaneously, beginning Week 0 of Maintenance study through Week 44.
  Interventions: Drug: Placebo SC
- Maintenance Study - Ustekinumab 90mg SC every 12 weeks (Experimental): Participants in clinical response (at Week 8 or Week 16) to Induction treatment with single IV infusion of Ustekinumab will be randomized to receive ustekinumab 90 mg subcutaneously every 12 weeks, beginning Week 0 of Maintenance study through Week 44.
  Interventions: Drug: Ustekinumab SC
- Maintenance Study - Ustekinumab 90mg SC every 8 weeks (q8w) (Experimental): Participants in clinical response (at Week 8 or Week 16) to Induction treatment with single IV infusion of Ustekinumab will be randomized to receive ustekinumab 90 mg subcutaneously every 8 weeks, beginning Week 0 of Maintenance study through Week 44.
  Interventions: Drug: Ustekinumab SC
- Maintenance Study - Placebo IV - Responder - Placebo SC (Other): Participants in clinical response to Induction treatment with IV Placebo will receive placebo subcutaneously, beginning Week 0 of Maintenance study through Week 44. Participants are not randomized.
  Interventions: Drug: Placebo SC
- Maintenance Study-Delayed Responder-Ustekinumab 90mg SC q8w (Other): Participants without clinical response to induction treatment ustekinumab (130 mg or 6 mg/kg [IV]) at Week 8 but in clinical response at Week 16 after receiving Induction Ustekinumab at week 8 (delayed responders) will receive ustekinumab 90 mg subcutaneously every 8 weeks, beginning Week 0 of Maintenance study through Week 44. Participants are not randomized.
  Interventions: Drug: Ustekinumab SC

INTERVENTIONS:
Drug: Placebo IV — Placebo will be administered as intravenous infusion.
  Arms: Induction Study - Placebo Intravenous (IV); Induction study-Ustekinumab Nonresponders at Week 8
Drug: Placebo SC — Placebo will be administered Subcutaneously.
  Arms: Induction Study- Placebo- Nonresponsders at Week 8; Maintenance Study - Placebo IV - Responder - Placebo SC; Maintenance Study - Placebo Subcutaneous (SC)
Drug: Ustekinumab IV — Ustekinumab will be administered as intravenous infusion at Week 0 or Week 8 in Induction Study.
  Arms: Induction Study - Ustekinumab 130 milligram (mg) IV; Induction Study - Ustekinumab 6 mg/kg IV; Induction Study- Placebo- Nonresponsders at Week 8
Drug: Ustekinumab SC — Ustekinumab will be administered as subcutaneously.
  Arms: Induction study-Ustekinumab Nonresponders at Week 8; Maintenance Study - Ustekinumab 90mg SC every 12 weeks; Maintenance Study - Ustekinumab 90mg SC every 8 weeks (q8w); Maintenance Study-Delayed Responder-Ustekinumab 90mg SC q8w

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ustekinumab as intravenous (IV: into the vein) infusion in induction study in participants with moderately to severely active Ulcerative Colitis (UC) and as subcutaneous (SC) administration in maintenance study in participants with moderately to severely active Ulcerative Colitis (UC) who have demonstrated a clinical response to Induction treatment with IV ustekinumab.

DETAILED DESCRIPTION:
This is a Phase 3, randomized (assignment of study drug by chance), double-blind (neither the participant or study staff will know the identity of study drugs), placebo-controlled (placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), parallel-group (a medical research study comparing the response in 2 or more groups of participants receiving different interventions), multi-center (more than one clinical site will work on a medical research study), protocol of ustekinumab. The protocol will consist of 2 studies: an Induction study and a Maintenance study with unique endpoints. Screening period will be up to 8 Weeks. Induction study will be at least 8 weeks duration for each participant. Participant with clinical response in the Induction study will be eligible for the Maintenance study. The Maintenance study will be 44 weeks duration. After completion of the maintenance study, a long term extension will follow eligible participants for an additional 3 years. Clinical remission will be evaluated at Week 8 in the Induction study. Clinical remission among ustekinumab Induction responders will be evaluated at week 44 in the Maintenance study. Participants' safety will be monitored throughout.

ELIGIBILITY:
Inclusion Criteria:

* Has a clinical diagnosis of Ulcerative Colitis (UC) at least 3 months before Screening
* Has moderately to severely active UC, defined as a Baseline (Week 0) Mayo score of 6 to 12, including a Screening endoscopy subscore of the Mayo score greater than or equal to (>=) 2 as determined by a central reading of the video endoscopy
* Have failed biologic therapy, that is, have received treatment with 1 or more tumour necrosis factor (TNF) antagonists or vedolizumab at a dose approved for the treatment of UC, and have a documented history of failure to respond to or tolerate such treatment; OR Be naïve to biologic therapy (TNF antagonists or vedolizumab) or have received biologic therapy but have not demonstrated a history of failure to respond to, or tolerate, a biologic therapy and have a prior or current UC medication history that includes at least 1 of the following: a. Inadequate response to or failure to tolerate current treatment with oral corticosteroids or immunomodulators (6-mercaptopurine [6-MP] or azathioprine [AZA]) OR b. History of failure to respond to, or tolerate, at least 1 of the following therapies: oral or IV corticosteroids or immunomodulators (6-MP or AZA) OR c. History of corticosteroid dependence (that is, an inability to successfully taper corticosteroids without a return of the symptoms of UC)
* Before the first administration of study agent, the following conditions must be met: vedolizumab must have been discontinued for at least 4 months and anti-tumor necrosis factors (TNFs) for at least 8 weeks

Exclusion Criteria:

* Has severe extensive colitis and is at imminent risk of colectomy
* Has UC limited to the rectum only or to < 20 centimeters (cm) of the colon
* Presence of a stoma or history of a fistula
* Participants with history of extensive colonic resection (for example, less than 30 cm of colon remaining) that would prevent adequate evaluation of the effect of study agent on clinical disease activity
* Participants with history of colonic mucosal dysplasia. Participants will not be excluded from the study because of a pathology finding of "indefinite dysplasia with reactive atypia''

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 961 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (247):
- United States (68):
  - Birmingham, Alabama
  - La Mirada, California
  - Los Angeles, California
  - Newport Beach, California
  - Torrance, California
  - Vallejo, California
  - Lone Tree, Colorado
  - Farmington, Connecticut
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Largo, Florida
  - Miami, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Macon, Georgia
  - Suwanee, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Evanston, Illinois
  - Urbana, Illinois
  - Indianapolis, Indiana
  - Pratt, Kansas
  - Crestview Hills, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Houma, Louisiana
  - Shreveport, Louisiana
  - Columbia, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Chesterfield, Michigan
  - Troy, Michigan
  - Ypsilanti, Michigan
  - Rochester, Minnesota
  - Jackson, Mississippi
  - Marlton, New Jersey
  - Morristown, New Jersey
  - Brooklyn, New York
  - Mineola, New York
  - New York, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - The Bronx, New York
  - Cincinnati, Ohio
  - Mentor, Ohio
  - Portland, Oregon
  - Doylestown, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Sayre, Pennsylvania
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Irving, Texas
  - San Antonio, Texas
  - Southlake, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Chesapeake, Virginia
  - Fairfax, Virginia
  - Roanoke, Virginia
  - Seattle, Washington
- Australia (10):
  - Bedford
  - Clayton
  - Concord
  - Fitzroy
  - Five Dock
  - Garran
  - Heidelberg
  - Liverpool
  - Melbourne
  - South Brisbane
- Austria (2):
  - Salzburg
  - Vienna
- Belgium (6):
  - Antwerp
  - Ghent
  - Kortrijk
  - Leuven
  - Liège
  - Roeselaere
- Bulgaria (5):
  - Pleven
  - Rousse
  - Sevlievo
  - Sofia
  - Varna
- Canada (7):
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Brandon, Manitoba
  - Winnipeg, Manitoba
  - Greater Sudbury, Ontario
  - London, Ontario
  - Montreal, Quebec
- Czechia (3):
  - Hradec Králové
  - Pilsen
  - Prague
- Denmark (2):
  - Aarhus
  - Odense
- France (11):
  - Amiens
  - Bordeaux
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Pierre-Bénite
  - Reims
  - Rennes
  - Saint-Etienne
  - Toulouse
- Germany (10):
  - Berlin
  - Essen
  - Freiburg im Breisgau
  - Hanover
  - Kiel
  - Leipzig
  - Lüneburg
  - Mannheim
  - Minden
  - Münster
- Hungary (10):
  - Balatonfüred
  - Békéscsaba
  - Budapest
  - Debrecen
  - Miskolc
  - Mosonmagyaróvár
  - Szekszárd
  - Székesfehérvár
  - Szombathely
  - Vác
- Israel (9):
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Petach Tikvah
  - Tel Aviv
  - Tel Litwinsky
- Japan (42):
  - Ageo-shi
  - Asahikawa
  - Bunkyō City
  - Chiba
  - Chikushinoshi
  - Fujiidera
  - Fukuoka-ken
  - Higashi-Ibaraki
  - Hirosaki
  - Hiroshima
  - Isesaki
  - Izumo
  - Kagoshima
  - Kahoku
  - Kobe
  - Kochi
  - Kurume
  - Kyoto
  - Midori-ku
  - Nagasaki
  - Nara
  - Nishinomiya
  - Numakunai
  - Osaka
  - Ōita
  - Saga
  - Saga-ken
  - Saitama
  - Sakura
  - Sapporo
  - Sendai
  - Shizuoka
  - Sunto-gun
  - Takamatsu
  - Tokorozawa
  - Tokyo
  - Toyama
  - Toyota
  - Tsu
  - Tsuchiura
  - Wakayama
  - Yamanashi
- Netherlands (2):
  - Amsterdam
  - Maastricht
- New Zealand (5):
  - Auckland
  - Christchurch
  - Dunedin
  - Lower Hutt
  - Milford
- Poland (8):
  - Gdansk
  - Krakow
  - Lodz
  - Puławy
  - Sopot
  - Szczecin
  - Warsaw
  - Wroclaw
- Romania (4):
  - Bucharest
  - Oradea
  - Romania
  - Timișoara
- Russia (10):
  - Irkutsk
  - Kazan'
  - Moscow
  - Moscva
  - Novosibirsk
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Stavropol
  - Ufa
- Serbia (4):
  - Belgrade
  - Kragujevac
  - Niš
  - Vojvodina
- Slovakia (2):
  - Bratislava
  - Prešov
- South Korea (4):
  - Daegu
  - Guri-si
  - Seoul
  - Suwon
- Ukraine (13):
  - Chernivtsi
  - Dnipropetrovsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiyv
  - Kyiv
  - Lviv
  - Odesa
  - Sumy
  - Uzhhorod
  - Vinnytsia
  - Zaporizhzhia
  - Zhaporozhia
- United Kingdom (10):
  - Birmingham
  - Cambridge
  - Coventry
  - Doncaster
  - Edinburgh
  - Liverpool
  - London
  - Salford
  - Southampton
  - Sutton in Ashfield

REFERENCES:
- [Derived] Danese S, Leong RW, Sands BE, Ma T, Marano C, Peyrin-Biroulet L. Clinical Trial: Association Between Early Disease Clearance and Long-Term Outcomes-4-Year Results From the Phase 3 UNIFI Study of Ustekinumab in Ulcerative Colitis. Aliment Pharmacol Ther. 2025 Sep;62(5):483-492. doi: 10.1111/apt.70264. Epub 2025 Jul 16. PMID 40668079
- [Derived] Solitano V, Panaccione R, Sands BE, Wang Z, Hogan M, Zou G, Peyrin-Biroulet L, Danese S, Cornfield LJ, Feagan BG, Singh S, Jairath V, Ma C. Responsiveness of different disease activity indices in moderate-to-severe ulcerative colitis. Med. 2025 Feb 14;6(2):100512. doi: 10.1016/j.medj.2024.09.001. Epub 2024 Oct 4. PMID 39368474
- [Derived] Ghosh S, Feagan BG, Ott E, Gasink C, Godwin B, Marano C, Miao Y, Ma T, Loftus EV Jr, Sandborn WJ, Danese S, Abreu MT, Sands BE. Safety of Ustekinumab in Inflammatory Bowel Disease: Pooled Safety Analysis Through 5 Years in Crohn's Disease and 4 Years in Ulcerative Colitis. J Crohns Colitis. 2024 Aug 6;18(7):1091-1101. doi: 10.1093/ecco-jcc/jjae013. PMID 38310565
- [Derived] Afif W, Arasaradnam RP, Abreu MT, Danese S, Sandborn WJ, Miao Y, Zhang H, Panaccione R, Hisamatsu T, Scherl EJ, Leong RW, Rowbotham DS, Peyrin-Biroulet L, Sands BE, Marano C. Efficacy and Safety of Ustekinumab for Ulcerative Colitis Through 4 Years: Final Results of the UNIFI Long-Term Maintenance Study. Am J Gastroenterol. 2024 May 1;119(5):910-921. doi: 10.14309/ajg.0000000000002621. Epub 2023 Dec 14. PMID 38095692
- [Derived] Chen R, Li L, Tie Y, Chen M, Zhang S. Trajectory of fecal lactoferrin for predicting prognosis in ulcerative colitis. Precis Clin Med. 2023 Sep 5;6(3):pbad022. doi: 10.1093/pcmedi/pbad022. eCollection 2023 Sep. PMID 38025971
- [Derived] Danese S, Sands BE, Abreu MT, O'Brien CD, Bravata I, Nazar M, Miao Y, Wang Y, Rowbotham D, Leong RWL, Arasaradnam RP, Afif W, Marano C. Early Symptomatic Improvement After Ustekinumab Therapy in Patients With Ulcerative Colitis: 16-Week Data From the UNIFI Trial. Clin Gastroenterol Hepatol. 2022 Dec;20(12):2858-2867.e5. doi: 10.1016/j.cgh.2022.02.050. Epub 2022 Mar 8. PMID 35276329
- [Derived] Panaccione R, Danese S, Sandborn WJ, O'Brien CD, Zhou Y, Zhang H, Adedokun OJ, Tikhonov I, Targan S, Abreu MT, Hisamatsu T, Scherl EJ, Leong RW, Rowbotham DS, Arasaradnam RP, Sands BE, Marano C. Ustekinumab is effective and safe for ulcerative colitis through 2 years of maintenance therapy. Aliment Pharmacol Ther. 2020 Dec;52(11-12):1658-1675. doi: 10.1111/apt.16119. Epub 2020 Oct 21. PMID 33086438
- [Derived] Sandborn WJ, Feagan BG, Danese S, O'Brien CD, Ott E, Marano C, Baker T, Zhou Y, Volger S, Tikhonov I, Gasink C, Sands BE, Ghosh S. Safety of Ustekinumab in Inflammatory Bowel Disease: Pooled Safety Analysis of Results from Phase 2/3 Studies. Inflamm Bowel Dis. 2021 Jun 15;27(7):994-1007. doi: 10.1093/ibd/izaa236. PMID 32964215
- [Derived] Li K, Marano C, Zhang H, Yang F, Sandborn WJ, Sands BE, Feagan BG, Rubin DT, Peyrin-Biroulet L, Friedman JR, De Hertogh G. Relationship Between Combined Histologic and Endoscopic Endpoints and Efficacy of Ustekinumab Treatment in Patients With Ulcerative Colitis. Gastroenterology. 2020 Dec;159(6):2052-2064. doi: 10.1053/j.gastro.2020.08.037. Epub 2020 Aug 25. PMID 32853634
- [Derived] Sands BE, Sandborn WJ, Panaccione R, O'Brien CD, Zhang H, Johanns J, Adedokun OJ, Li K, Peyrin-Biroulet L, Van Assche G, Danese S, Targan S, Abreu MT, Hisamatsu T, Szapary P, Marano C; UNIFI Study Group. Ustekinumab as Induction and Maintenance Therapy for Ulcerative Colitis. N Engl J Med. 2019 Sep 26;381(13):1201-1214. doi: 10.1056/NEJMoa1900750. PMID 31553833

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction Study(IS): Placebo Intravenous (IV): Participants received single dose of placebo as intravenous (IV) infusion at Week 0. Participants with clinical response at Week (W) 8 were eligible to enter the maintenance study. Participants who did not achieve clinical response at Week 8 received weight-range based dose of ustekinumab approximating 6 mg/kg IV + placebo SC at Week 8. At Week 16, participants who did not achieve clinical response at Week 8 were re-evaluated for clinical response. Participants with clinical response at Week 16 were eligible to enter the maintenance study. Participants who did not achieve clinical response at Week 16 were not eligible to enter the maintenance study and had a safety follow-up visit up to 20 weeks after their last dose of study agent.
- IS: Ustekinumab 130 Milligram (mg) IV: Participants received single dose of ustekinumab 130 mg as IV infusion at Week 0. Participants with clinical response at Week 8 were eligible to enter the maintenance study. Participants who did not achieve clinical response at Week 8 received 1 dose of ustekinumab 90 mg SC+ placebo IV at Week 8. At Week 16, participants who did not achieve clinical response at Week 8 were re-evaluated for clinical response. Participants with clinical response at Week 16 were eligible to enter the maintenance study. Participants who did not achieve clinical response at Week 16 were not eligible to enter the maintenance study and had a safety follow-up visit up to 20 weeks after their last dose of study agent.
- IS: Ustekinumab Approximately 6mg/kg IV: Participants received weight range based dose of ustekinumab approximating 6 milligram per kilogram (mg/kg) (ustekinumab 260 mg [body weight <=55 kg], 390 mg [body weight >55 kg but ≤85 kg] and 520 mg [body weight >85 kg]), as IV infusion at Week 0. Participants with clinical response at Week 8 were eligible to enter the maintenance study. Participants who did not achieve clinical response at Week 8 received 1 dose of ustekinumab 90 mg SC+ placebo IV at Week 8. At Week 16, participants who did not achieve clinical response at Week 8 were re-evaluated for clinical response. Participants with clinical response at Week 16 were eligible to enter the maintenance study. Participants who did not achieve clinical response at Week 16 were not eligible to enter the maintenance study and had a safety follow-up visit up to 20 weeks after their last dose of study agent.
- Maintenance Study(MS): Placebo Subcutaneous (SC): Participants in clinical response (at Week 8 or Week 16) to Induction treatment with single IV infusion of Ustekinumab who were randomized to receive placebo subcutaneously, beginning Week 0 of Maintenance study through Week 44.
- MS: Ustekinumab 90mg SC Every 12 Weeks (q12w): Participants who were randomized to receive ustekinumab (ie, 130 mg IV or approximately 6 mg/kg IV) at Week 0 of the induction study and were in clinical response at induction Week 8 and participants who were randomized to receive placebo at Week 0 of the induction study and were not in clinical response at induction Week 8 but were in clinical response at induction Week 16 after receiving a dose of IV ustekinumab (approximately 6 mg/kg) at induction Week 8 (placebo to ustekinumab 6 mg/kg IV) were randomized to receive ustekinumab 90 mg SC every 12 weeks (q12w) beginning at Week 0 of maintenance study through Week 44.
- MS: Ustekinumab 90mg SC Every 8 Weeks (q8w): Participants who were randomized to receive ustekinumab (ie, 130 mg IV or approximately 6 mg/kg IV) at Week 0 of the induction study and were in clinical response at induction Week 8 and participants who were randomized to receive placebo at Week 0 of the induction study and were not in clinical response at induction Week 8 but were in clinical response at induction Week 16 after receiving a dose of IV ustekinumab (approximately 6 mg/kg) at induction Week 8 (placebo to ustekinumab 6 mg/kg IV) were randomized to receive ustekinumab 90 mg SC every 8 weeks (q8w), beginning at Week 0 of maintenance study through Week 44.
- MS: Placebo IV (IS - Responders) to Placebo SC: Participants with clinical response to Induction Week 0 treatment with placebo IV received placebo SC, beginning at Week 0 of maintenance study through Week 44 (non-randomized participants).
- MS: Ustekinumab Delayed Responders(IS) to UST 90mg SC q8w: Participants who were delayed responders to ustekinumab induction (were not in clinical response to induction treatment ustekinumab (130 mg or approximately 6 mg/kg [IV]) at Week 8 but were in clinical response at Week 16, after receiving ustekinumab 90 mg SC at Week 8) and received ustekinumab 90 mg SC every 8 weeks, beginning at Week 0 of maintenance study through Week 44 (non-randomized participants).
- Long Term Extension (LTE): Placebo SC: Participants who were randomized to receive placebo SC in the maintenance study and received placebo SC at the first dosing visit (Week 48) of long term extension (LTE).
- LTE: Ustekinumab 90 mg SC q12w: Participants who were randomized to receive ustekinumab 90 mg SC every 12 weeks (q12w) in the maintenance study and received ustekinumab 90 mg SC at the first dosing visit (Week 48) of the LTE.
- LTE: Ustekinumab 90 mg SC q8w: Participants who were randomized to receive ustekinumab 90 mg SC every 8 weeks (q8w) in the maintenance study and received ustekinumab 90 mg SC at the first dosing visit (Week 48) of the LTE.
- LTE: Placebo IV (IS - Responders) to Placebo SC: Participants with clinical response to Induction Week 0 treatment with placebo IV received placebo SC in the maintenance study and the LTE through Week 200 (non-randomized participants).
- LTE: Ustekinumab Delayed Responders (IS) to UST 90mg SC q8w: Participants who were delayed responders to ustekinumab induction (were not in clinical response to induction treatment ustekinumab (130 mg or approximately 6 mg/kg [IV]) at Week 8 but were in clinical response at Week 16, after receiving ustekinumab 90 mg SC at Week 8) and received ustekinumab 90 mg SC q8w in the maintenance study and the LTE through Week 200 (non-randomized participants).
Period: Induction Study (8 Weeks)
Arm/Group | Induction Study(IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6mg/kg IV | Maintenance Study(MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90mg SC Every 8 Weeks (q8w) | MS: Placebo IV (IS - Responders) to Placebo SC | MS: Ustekinumab Delayed Responders(IS) to UST 90mg SC q8w | Long Term Extension (LTE): Placebo SC | LTE: Ustekinumab 90 mg SC q12w | LTE: Ustekinumab 90 mg SC q8w | LTE: Placebo IV (IS - Responders) to Placebo SC | LTE: Ustekinumab Delayed Responders (IS) to UST 90mg SC q8w
Started | 319 | 320 | 322 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 296 | 309 | 307 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 23 | 11 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 17 | 9 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Study (44 Weeks)
Arm/Group | Induction Study(IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6mg/kg IV | Maintenance Study(MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90mg SC Every 8 Weeks (q8w) | MS: Placebo IV (IS - Responders) to Placebo SC | MS: Ustekinumab Delayed Responders(IS) to UST 90mg SC q8w | Long Term Extension (LTE): Placebo SC | LTE: Ustekinumab 90 mg SC q12w | LTE: Ustekinumab 90 mg SC q8w | LTE: Placebo IV (IS - Responders) to Placebo SC | LTE: Ustekinumab Delayed Responders (IS) to UST 90mg SC q8w
Started | 0 | 0 | 0 | 175 | 172 | 176 | 103 | 157 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 132 | 148 | 158 | 76 | 128 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 43 | 24 | 18 | 27 | 29 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 19 | 8 | 4 | 11 | 10 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 19 | 9 | 6 | 12 | 12 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 5 | 7 | 8 | 4 | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Long-term Extension Period (176 Weeks)
Arm/Group | Induction Study(IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6mg/kg IV | Maintenance Study(MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90mg SC Every 8 Weeks (q8w) | MS: Placebo IV (IS - Responders) to Placebo SC | MS: Ustekinumab Delayed Responders(IS) to UST 90mg SC q8w | Long Term Extension (LTE): Placebo SC | LTE: Ustekinumab 90 mg SC q12w | LTE: Ustekinumab 90 mg SC q8w | LTE: Placebo IV (IS - Responders) to Placebo SC | LTE: Ustekinumab Delayed Responders (IS) to UST 90mg SC q8w
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 115 | 141 | 143 | 73 | 116
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 99 | 101 | 0 | 95
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 81 | 42 | 42 | 73 | 21
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 17 | 10 | 11 | 9
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 6 | 12 | 7 | 6
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63 | 19 | 19 | 55 | 6

BASELINE CHARACTERISTICS:
Population: The primary efficacy analysis set consisted of all participants randomized in the study.
Groups:
- Induction Study (IS): Placebo Intravenous (IV): Participants received single dose of placebo as intravenous (IV) infusion at Week 0. Participants with clinical response at Week (W) 8 were eligible to enter the maintenance study. Participants who did not achieve clinical response at Week 8 received weight-range based dose of ustekinumab approximating 6 mg/kg IV + placebo SC at Week 8. At Week 16, participants who did not achieve clinical response at Week 8 were re-evaluated for clinical response. Participants with clinical response at Week 16 were eligible to enter the maintenance study. Participants who did not achieve clinical response at Week 16 were not eligible to enter the maintenance study and had a safety follow-up visit up to 20 weeks after their last dose of study agent.
- IS: Ustekinumab 130 Milligram (mg) IV: Participants received single dose of ustekinumab 130 mg as IV infusion at Week 0. Participants with clinical response at Week 8 were eligible to enter the maintenance study. Participants who did not achieve clinical response at Week 8 received 1 dose of ustekinumab 90 mg SC+ placebo IV at Week 8. At Week 16, participants who did not achieve clinical response at Week 8 were re-evaluated for clinical response. Participants with clinical response at Week 16 were eligible to enter the maintenance study. Participants who did not achieve clinical response at Week 16 were not eligible to enter the maintenance study and had a safety follow-up visit up to 20 weeks after their last dose of study agent.Participants received single dose of ustekinumab 130 mg as IV infusion at Week 0. Participants with clinical response at Week 8 were eligible to enter the maintenance study. Participants who did not achieve clinical response at Week 8 received 1 dose of ustekinumab 90 mg SC+ placebo IV at Week 8. At Week 16, participants who did not achieve clinical response at Week 8 were re-evaluated for clinical response. Participants with clinical response at Week 16 were eligible to enter the maintenance study. Participants who did not achieve clinical response at Week 16 were not eligible to enter the maintenance study and had a safety follow-up visit up to 20 weeks after their last dose of study agent.
- Total: Total of all reporting groups
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6mg/kg IV | Maintenance Study(MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90mg SC Every 8 Weeks (q8w) | MS: Placebo IV (IS - Responders) to Placebo SC | MS: Ustekinumab Delayed Responders(IS) to UST 90mg SC q8w | Long Term Extension (LTE): Placebo SC | LTE: Ustekinumab 90 mg SC q12w | LTE: Ustekinumab 90 mg SC q8w | LTE: Placebo IV (IS - Responders) to Placebo SC | LTE: Ustekinumab Delayed Responders (IS) to UST 90mg SC q8w | Total
Number analyzed (Participants) | 319 | 320 | 322 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 961
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (13.50) | 42.2 (13.94) | 41.7 (13.67) |  |  |  |  |  |  |  |  |  |  | 41.7 (13.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 130 | 127 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 379
  Male | 197 | 190 | 195 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 582
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24
  Not Hispanic or Latino | 292 | 295 | 290 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 877
  Unknown or Not Reported | 17 | 18 | 25 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 60
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 1 |  |  |  |  |  |  |  |  |  |  | 1
  Asian | 48 | 46 | 49 |  |  |  |  |  |  |  |  |  |  | 143
  Black or African American | 3 | 6 | 0 |  |  |  |  |  |  |  |  |  |  | 9
  Other | 8 | 9 | 12 |  |  |  |  |  |  |  |  |  |  | 29
  White | 248 | 239 | 243 |  |  |  |  |  |  |  |  |  |  | 730
  Unknown or Not Reported | 12 | 20 | 17 |  |  |  |  |  |  |  |  |  |  | 49
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 7 | 8 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26
  Austria | 0 | 2 | 2 |  |  |  |  |  |  |  |  |  |  | 4
  Belgium | 22 | 10 | 7 |  |  |  |  |  |  |  |  |  |  | 39
  Bulgaria | 8 | 9 | 4 |  |  |  |  |  |  |  |  |  |  | 21
  Canada | 7 | 6 | 3 |  |  |  |  |  |  |  |  |  |  | 16
  Czech Republic | 8 | 9 | 13 |  |  |  |  |  |  |  |  |  | 0 | 30
  Denmark | 0 | 0 | 2 |  |  |  |  |  |  |  |  |  |  | 2
  France | 14 | 21 | 19 |  |  |  |  |  |  |  |  |  |  | 54
  Germany | 19 | 14 | 12 |  |  |  |  |  |  |  |  |  |  | 45
  Hungary | 11 | 12 | 16 | 0 |  |  |  |  |  |  |  |  |  | 39
  Israel | 0 | 3 | 3 | 0 |  |  |  |  |  |  |  |  |  | 6
  Italy | 10 | 11 | 12 |  |  |  |  |  |  |  |  |  |  | 33
  Japan | 34 | 34 | 39 |  |  |  |  |  |  |  |  |  |  | 107
  Netherlands | 5 | 8 | 3 |  |  |  |  |  |  |  |  |  |  | 16
  New Zealand | 4 | 4 | 11 |  |  |  |  |  |  |  |  |  |  | 19
  Poland | 25 | 26 | 20 |  |  |  |  |  |  |  |  |  |  | 71
  Romania | 7 | 9 | 8 |  |  |  |  |  |  |  |  |  |  | 24
  Russia | 26 | 22 | 26 |  |  |  |  |  |  |  |  |  |  | 74
  Serbia | 1 | 6 | 3 |  |  |  |  |  |  |  |  |  |  | 10
  Slovakia | 4 | 4 | 2 |  |  |  |  |  |  |  |  |  |  | 10
  Ukraine | 32 | 26 | 31 |  |  |  |  |  |  |  |  |  |  | 89
  United Kingdom | 5 | 3 | 13 |  |  |  |  |  |  |  |  |  |  | 21
  United States | 60 | 63 | 56 |  |  |  |  |  |  |  |  |  |  | 179
  Korea | 10 | 10 | 6 |  |  |  |  |  |  |  |  |  |  | 26

OUTCOME MEASURES:

1. Primary Outcome: Induction Study - Number of Participants With Clinical Remission at Week 8 (As Per Global Definition)
Description: As per global definition, clinical remission is defined as a Mayo score less than or equal to (<=)2 points, with no individual subscore greater than (>)1. The Mayo score consists of 4 subscores (stool frequency, rectal bleeding [RB], endoscopy findings, and physician's global assessment [PGA]), rated as 0 (normal) to 3 (severe). Total score was calculated as the sum of 4 subscores and values range from 0 to 12 scores, where 3 to 5 = mild; 6 to 10 = moderate; and 11 to 12 = severe; higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant ulcerative colitis (UC) medication or an ostomy or colectomy prior to the Week 8 or who had all 4 Mayo subscores missing at Week 8 were considered not to be in clinical remission. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 8
Population: The primary efficacy analysis set (PEAS) consisted of all participants randomized in the induction study.
Measure: Count of Participants; unit: Participants
Groups:
- IS: Ustekinumab Approximately 6 mg/kg IV: Participants received weight range based dose of ustekinumab approximating 6 milligram per kilogram (mg/kg) (ustekinumab 260 mg [body weight <=55 kg], 390 mg [body weight >55 kg but ≤85 kg] and 520 mg [body weight >85 kg]), as IV infusion at Week 0. Participants with clinical response at Week 8 were eligible to enter the maintenance study. Participants who did not achieve clinical response at Week 8 received 1 dose of ustekinumab 90 mg SC+ placebo IV at Week 8. At Week 16, participants who did not achieve clinical response at Week 8 were re-evaluated for clinical response. Participants with clinical response at Week 16 were eligible to enter the maintenance study. Participants who did not achieve clinical response at Week 16 were not eligible to enter the maintenance study and had a safety follow-up visit up to 20 weeks after their last dose of study agent.
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants | 17 | 50 | 50
Statistical Analysis 1: Comparison: Induction Study (IS): Placebo Intravenous (IV) vs IS: Ustekinumab 130 Milligram (mg) IV; Statistical Analysis 1; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted treatment difference = 10.3, 95% CI 2-sided [5.7 to 14.9] — Treatment difference between ustekinumab group and placebo group was adjusted with Cochran-Mantel-Haenszel (CMH) weight
Statistical Analysis 2: Comparison: Induction Study (IS): Placebo Intravenous (IV) vs IS: Ustekinumab Approximately 6 mg/kg IV; Statistical Analysis 2; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted treatment difference = 10.2, 95% CI 2-sided [5.6 to 14.8] — Treatment difference between ustekinumab group and placebo group was adjusted with Cochran-Mantel-Haenszel (CMH) weight

2. Primary Outcome: Induction Study - Number of Participants With Clinical Remission at Week 8 (As Per US Definition)
Description: As per US definition, clinical remission was defined as absolute stool number <=3, a Mayo rectal bleeding subscore of 0 (no blood seen), and a Mayo endoscopy subscore of 0 (normal or inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]) without the physician's global assessment. Absolute stool number is average of daily stool number over the three days. The Mayo rectal bleeding and endoscopy findings subscores were rated as 0 (normal) to 3 (severe). Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 or who were missing all 3 of the Mayo components pertaining to this outcome measure (OM) (absolute stool number, rectal bleeding subscore, and Mayo endoscopy subscore) at Week 8 were considered not to be in clinical remission. Endoscopy subscore as assessed during central review of the video of the endoscopy was used.
Time Frame: Week 8
Population: PEAS consisted of all participants randomized in the induction study.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants | 20 | 53 | 61
Statistical Analysis 1: Comparison: Induction Study (IS): Placebo Intravenous (IV) vs IS: Ustekinumab 130 Milligram (mg) IV; Statistical Analysis 1; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted treatment difference = 10.3, 97.5% CI 2-sided [4.8 to 15.8] — Treatment difference between ustekinumab group and placebo group was adjusted with Cochran-Mantel-Haenszel (CMH) weight
Statistical Analysis 2: Comparison: Induction Study (IS): Placebo Intravenous (IV) vs IS: Ustekinumab Approximately 6 mg/kg IV; Statistical Analysis 2; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted treatment difference = 12.7, 97.5% CI 2-sided [7.0 to 18.4] — Treatment difference between ustekinumab group and placebo group was adjusted with Cochran-Mantel-Haenszel (CMH) weight

3. Primary Outcome: Maintenance Study: Number of Participants With Clinical Remission at Week 44 (As Per Global Definition)
Description: As per global definition, clinical remission was defined as a Mayo score <=2 points, with no individual subscore >1. The Mayo score consists of 4 subscores (stool frequency, rectal bleeding, endoscopy findings, and physician's global assessment), rated as 0 (normal) to 3 (severe). Total score was calculated as the sum of 4 subscores and values range from 0 to 12 scores, where 3 to 5 = mild; 6 to 10 = moderate; and 11 to 12 = severe; higher scores indicate worsening of the disease. Participants who had a prohibited change in UC medication or an ostomy or colectomy or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 or who had all 4 Mayo subscores missing at Week 44 were considered not to be in clinical remission. Endoscopy subscore as assessed during central review of the video of the endoscopy was used.
Time Frame: Week 44
Population: PEAS consisted of all participants who were in clinical response to IV ustekinumab induction and were randomized at Week 0 of the maintenance study to ustekinumab 90 mg SC every 8 weeks (q8w), ustekinumab 90 mg SC every 12 weeks (q12w), or placebo SC.
Measure: Count of Participants; unit: Participants
Groups:
- Maintenance Study (MS): Placebo Subcutaneous (SC): Participants who were randomized to receive ustekinumab (i.e., 130 mg IV or approximately 6 mg/kg IV) at Week 0 of the induction study and were in clinical response at induction Week 8 and participants who were randomized to receive placebo at Week 0 of the induction study and were not in clinical response at induction Week 8 but were in clinical response at induction Week 16 after receiving a dose of IV ustekinumab (approximately 6 mg/kg) at induction Week 8 (placebo to ustekinumab 6 mg/kg IV) were randomized to receive placebo subcutaneous (SC), beginning at Week 0 of maintenance study through Week 44.
- MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w): Participants who were randomized to receive ustekinumab (ie, 130 mg IV or approximately 6 mg/kg IV) at Week 0 of the induction study and were in clinical response at induction Week 8 and participants who were randomized to receive placebo at Week 0 of the induction study and were not in clinical response at induction Week 8 but were in clinical response at induction Week 16 after receiving a dose of IV ustekinumab (approximately 6 mg/kg) at induction Week 8 (placebo to ustekinumab 6 mg/kg IV) were randomized to receive ustekinumab 90 mg SC every 12 weeks (q12w) beginning at Week 0 of maintenance study through Week 44.
- MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w): Participants who were randomized to receive ustekinumab (ie, 130 mg IV or approximately 6 mg/kg IV) at Week 0 of the induction study and were in clinical response at induction Week 8 and participants who were randomized to receive placebo at Week 0 of the induction study and were not in clinical response at induction Week 8 but were in clinical response at induction Week 16 after receiving a dose of IV ustekinumab (approximately 6 mg/kg) at induction Week 8 (placebo to ustekinumab 6 mg/kg IV) were randomized to receive ustekinumab 90 mg SC every 8 weeks (q8w), beginning at Week 0 of maintenance study through Week 44.
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants | 42 | 66 | 77
Statistical Analysis 1: Comparison: Maintenance Study (MS): Placebo Subcutaneous (SC) vs MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w); Statistical Analysis 1; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Adjusted treatment difference = 14.5, 95% CI 2-sided [5.5 to 23.6] — Treatment difference between ustekinumab group and placebo group was adjusted with CMH weight
Statistical Analysis 2: Comparison: Maintenance Study (MS): Placebo Subcutaneous (SC) vs MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w); Statistical Analysis 2; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted treatment difference = 19.7, 95% CI 2-sided [10.3 to 29.0] — Treatment difference between ustekinumab group and placebo group was adjusted with CMH weight

4. Primary Outcome: Maintenance Study: Number of Participants With Clinical Remission at Week 44 (as Per US Definition)
Description: Per US definition, clinical remission: absolute stool number <=3, a Mayo rectal bleeding subscore of 0 (no blood seen), and a Mayo endoscopy subscore of 0 (normal or inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]), without the physician's global assessment. Absolute stool number is average of daily stool number over the three days. The Mayo rectal bleeding and endoscopy findings subscores were rated as 0 (normal) to 3 (severe). Participants who had prohibited change in UC medication/ ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study agent due to lack of therapeutic effect/ due to AE of worsening of UC prior to Week 44 and who were missing all 3 of Mayo components pertaining to this OM (absolute stool number, rectal bleeding subscore, and Mayo endoscopy subscore) at Week 44 were considered not to be in clinical remission. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 44
Population: PEAS consisted of all participants who were in clinical response to IV ustekinumab induction and were randomized at Week 0 of the maintenance study to ustekinumab 90 mg SC q8w, ustekinumab 90 mg SC q12w, or placebo SC.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants | 43 | 68 | 75
Statistical Analysis 1: Comparison: Maintenance Study (MS): Placebo Subcutaneous (SC) vs MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w); Statistical Analysis 1; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Adjusted treatment difference = 15.1, 95% CI 2-sided [6.0 to 24.2] — Treatment difference between ustekinumab group and placebo group was adjusted with CMH weight
Statistical Analysis 2: Comparison: Maintenance Study (MS): Placebo Subcutaneous (SC) vs MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w); Statistical Analysis 2; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted treatment difference = 17.9, 95% CI 2-sided [8.6 to 27.2] — Treatment difference between ustekinumab group and placebo group was adjusted with CMH weight

5. Secondary Outcome: Induction Study: Number of Participants With Endoscopic Healing at Week 8
Description: Endoscopic healing is improvement in the endoscopic appearance of the mucosa. It is defined as Mayo endoscopic subscore = 0 (normal or inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]). Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 or who had a missing endoscopy score at Week 8 were considered not to have endoscopic healing. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 8
Population: PEAS consisted of all participants randomized in the induction study.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants | 44 | 84 | 87

6. Secondary Outcome: Induction Study: Number of Participants With Clinical Response at Week 8
Description: Clinical response was defined as a decrease from induction baseline in the Mayo score by >=30 percent (%) and >= 3 points, with either a decrease from baseline in the rectal bleeding subscore >=1 or a rectal bleeding subscore of 0 or 1. The Mayo score consists of 4 subscores (stool frequency, rectal bleeding, endoscopy findings, and physician's global assessment), rated as 0 (normal) to 3 (severe). Total score was calculated as the sum of 4 subscores and values range from 0 to 12 scores, where 3 to 5 = mild; 6 to 10 = moderate; and 11 to 12 = severe; higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 or who had all 4 Mayo subscores missing at Week 8 were considered not to be in clinical response. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 8
Population: PEAS consisted of all participants randomized in the induction study.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants | 100 | 164 | 199

7. Secondary Outcome: Induction Study - Change From Baseline in Total Inflammatory Bowel Disease Questionnaire (IBDQ) Score at Week 8
Description: The IBDQ is 32-item questionnaire for participants with Inflammatory Bowel Disease (IBD) used to evaluate disease-specific health-related quality of life. IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). The 32 items were grouped into 4 domains: bowel function, emotional status, systemic symptoms and social function. The 4 domains were scored as follows: 10 to 70 (bowel symptoms); 5 to 35 (systemic symptoms); 12 to 84 (emotional function); and 5 to 35 (social function). For each domain, higher score indicated better quality of life. Total score is sum of each item score and ranges from 32 to 224 with higher score indicating better quality of life. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 had their baseline value carried forward from the time of event onward or participants who had missing IBDQ score at Week 8 had their last value carried forward.
Time Frame: Baseline and Week 8
Population: PEAS consisted of all participants randomized in the induction study. Here, N (number of participants analyzed) signifies those participants who were analyzed for this outcome measure (OM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 317 | 316 | 321
Units on a scale | 16.1 (31.39) | 33.4 (32.53) | 35.0 (31.86)

8. Secondary Outcome: Maintenance Study: Number of Participants With Clinical Response up to Week 44
Description: Clinical response: decrease from induction baseline in Mayo score by >= 30% and >= 3 points, with either decrease from induction baseline in rectal bleeding subscore >=1 or rectal bleeding subscore of 0 or 1. Mayo score includes 4 subscores (stool frequency, rectal bleeding, endoscopy findings, physician's global assessment), rated as 0 (normal) to 3 (severe). Total score is sum of 4 subscores and values range from 0 to 12 scores, where 3 to 5= mild; 6 to 10= moderate; 11 to 12= severe; higher scores indicate worsening of disease. Participants who lost clinical response at any time before Week 44, had prohibited change in UC medication, ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study agent due to lack of therapeutic effect/ AE of worsening of UC before Week 44 or who had all 4 Mayo subscores missing at Week 44 were considered not to be in clinical response. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Up to Week 44
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants | 78 | 117 | 125

9. Secondary Outcome: Maintenance Study: Number of Participants With Endoscopic Healing at Week 44
Description: Endoscopic healing is improvement in the endoscopic appearance of the mucosa. It was defined as Mayo endoscopic subscore = 0 (normal or inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]). Participants who had prohibited change in UC medication, an ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study agent due to lack of therapeutic effect/ AE of worsening of UC prior to Week 44 or who had missing endoscopy score at Week 44 were considered not to have endoscopic healing. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 44
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants | 50 | 75 | 90

10. Secondary Outcome: Maintenance Study: Number of Participants With Clinical Remission and Not Receiving Concomitant Corticosteroids (Corticosteroid-free Clinical Remission) at Week 44 (As Per Global Definition)
Description: Per global definition, clinical remission was defined as Mayo score <=2 points, with no individual subscore >1. Mayo score consists of 4 subscores (stool frequency, rectal bleeding, endoscopy findings, and physician's global assessment), rated as 0 (normal) to 3 (severe). Total score: sum of 4 subscores and range from 0 to 12, where 3 to 5= mild; 6 to 10= moderate; and 11 to 12= severe; higher scores indicate worsening of disease. Participants who had prohibited change in UC medication/ ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study agent due to lack of therapeutic effect/ AE of worsening of UC before Week 44 or had all 4 Mayo subscores missing at Week 44 were considered not to have achieved OM of clinical remission and not receiving corticosteroids at Week 44. Participants who had missing value in corticosteroid use at Week 44 had their last value carried forward. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 44
Population: PEAS included all participants who were in clinical response to IV ustekinumab induction and were randomized at Week 0 of maintenance study to ustekinumab 90 mg SC q8w, ustekinumab 90 mg SC q12w/ placebo SC.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants | 41 | 65 | 74

11. Secondary Outcome: Maintenance Study: Number of Participants With Clinical Remission and Not Receiving Concomitant Corticosteroids (Corticosteroid-free Clinical Remission) at Week 44 (As Per US Definition)
Description: US definition of clinical remission: absolute stool number <=3, rectal bleeding subscore 0 (no blood seen), Mayo endoscopy subscore of 0(normal or inactive disease)/ 1 (mild disease [erythema, decreased vascular pattern, mild friability]). Absolute stool number: average of daily stool number over 3 days. Mayo rectal bleeding and endoscopy findings subscores rated: 0 (normal) to 3 (severe). Participants with prohibited change in UC medication/ostomy/colectomy/used rescue medication after clinical flare/ discontinued study agent due to lack of therapeutic effect/ AE of worsening of UC before Week 44 or were missing all 3 of Mayo components related to this OM (absolute stool number, rectal bleeding, and Mayo endoscopy subscore) at Week 44 were considered not in corticosteroid-free clinical remission at Week 44. Participants with missing value in corticosteroid use at Week 44 had last value carried forward. Endoscopy subscore assessed during central review of video of endoscopy was used.
Time Frame: Week 44
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants | 42 | 67 | 72

12. Secondary Outcome: Maintenance Study: Number of Participants With Clinical Remission up to Week 44 Among Participants Who Achieved Clinical Remission at Maintenance Study Baseline (As Per Global Definition)
Description: Global definition of clinical remission: Mayo score <=2 points, with no individual subscore >1. Mayo score includes 4 subscores (stool frequency, rectal bleeding, endoscopy findings, physician's global assessment), rated as 0 (normal) to 3 (severe). Total score: sum of 4 subscores and range from 0 to 12, where 3 to 5= mild; 6 to 10= moderate; and 11 to 12= severe; higher scores indicate worsening of disease. Participants who had prohibited change in UC medication/ ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study agent due to lack of therapeutic effect/ AE of worsening of UC before Week 44 or had all 4 Mayo subscores missing at Week 44 were considered not to be in clinical remission. Participants who were not in clinical remission at any time points when endoscopic scores were collected before Week 44 were considered not to be in clinical remission up to Week 44. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Up to Week 44
Population: PEAS consisted of all participants who were in clinical response to IV ustekinumab induction and were randomized at Week 0 of the maintenance study to ustekinumab 90 mg SC q8w, ustekinumab 90 mg SC q12w, or placebo SC, with participants who were in clinical remission at maintenance baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 45 | 40 | 38
Participants | 17 | 26 | 22

13. Secondary Outcome: Maintenance Study: Number of Participants With Clinical Remission up to Week 44 Among Participants Who Achieved Clinical Remission at Maintenance Study Baseline (As Per US Definition)
Description: US definition of clinical remission: absolute stool number <=3, Mayo rectal bleeding subscore of 0 (no blood seen), Mayo endoscopy subscore of 0 (normal/ inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]). Absolute stool number: average of daily stool number over 3 days. Mayo rectal bleeding and endoscopy subscores: 0 (normal) to 3 (severe). Participants with prohibited change in UC medication/ostomy/colectomy/used rescue medication after clinical flare/ discontinued study drug due to lack of therapeutic effect/ AE of worsening of UC before Week 44/ missing all 3 of Mayo components (absolute stool number, rectal bleeding, and Mayo endoscopy subscore) at Week 44 were considered not in clinical remission. Participants not in clinical remission at any time point when endoscopic scores collected before Week 44 considered not in clinical remission up to Week 44. Endoscopy subscore assessed during central review of video of endoscopy was used.
Time Frame: Up to Week 44
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 48 | 52 | 44
Participants | 16 | 32 | 27

14. Secondary Outcome: Induction Study - Number of Participants With Mucosal Healing at Week 8
Description: Mucosal healing is defined as having both endoscopic healing (EH) and histologic healing (HH). Endoscopic healing: an endoscopy subscore of 0 (normal or inactive disease) or 1 mild disease ([erythema, decreased vascular pattern, mild friability]). Histologic healing: neutrophil infiltration in <5% of crypts, no crypt destruction, and no erosions or ulcerations or granulation tissue. Participants who had prohibited change in concomitant UC medication/ ostomy/ colectomy before Week 8 or had missing endoscopy score/ were missing any component of histologic healing (that is assessment of neutrophils in crypts, crypt destruction/ erosions/ ulcerations/ granulations) at Week 8 or who had unevaluable biopsy (that is biopsy collected, but could not be assessed due to sample preparation or technical errors) at Week 8 but who did not achieve endoscopic healing, were considered not to have mucosal healing. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 8
Population: PEAS consisted of all participants randomized in the induction study, with participants whose mucosal healing status was determined at Week 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 316 | 316 | 315
Participants | 28 | 64 | 58

15. Secondary Outcome: Induction Study - Number of Participants in Clinical Remission With a Rectal Bleeding Subscore of 0 at Week 8 (As Per Global Definition)
Description: As per global definition, clinical remission is defined as Mayo score <=2 points, with no individual subscore >1. The Mayo score consists of 4 subscores (stool frequency, rectal bleeding, endoscopy findings, and physician's global assessment), rated as 0 (normal) to 3 (severe). Total score is calculated as sum of 4 subscores and values range from 0 to 12 scores, where 3 to 5 = mild; 6 to 10 = moderate; and 11 to 12 = severe; higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to Week 8 or who had missing rectal bleeding subscores at Week 8 were considered not to be in clinical remission with a rectal bleeding subscore of 0. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 8
Population: PEAS consisted of all participants randomized in the induction study.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants | 17 | 49 | 49

16. Secondary Outcome: Induction Study - Number of Participants in Symptomatic Remission at Week 8
Description: Symptomatic remission was defined as a Mayo stool frequency subscore of 0 (normal number of stools) or 1 (1-2 stools more than normal) and a rectal bleeding subscore of 0 (no blood seen). Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to Week 8 and/or both stool frequency and rectal bleeding subscores missing at Week 8 were considered not to be in symptomatic remission.
Time Frame: Week 8
Population: PEAS consisted of all participants randomized in the induction study.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants | 72 | 132 | 144

17. Secondary Outcome: Induction Study - Number of Participants in With Normal or Inactive Mucosal Disease at Week 8
Description: Normal or inactive mucosal disease is defined as an endoscopy score of 0. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to Week 8 or who had a missing endoscopy score at Week 8 were considered not to have normal or inactive mucosal disease. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 8
Population: PEAS consisted of all participants randomized in the induction study.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants | 12 | 33 | 25

18. Secondary Outcome: Induction Study - Change From Baseline in Mayo Score at Week 8
Description: The Mayo score consists of 4 subscores (stool frequency, rectal bleeding, endoscopy findings, and physician's global assessment), rated as 0 (normal) to 3 (severe). Total score is calculated as the sum of 4 subscores and values range from 0 to 12 scores, where 3 to 5 = mild; 6 to 10 = moderate; and 11 to 12 = severe; higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 had their baseline Mayo score carried forward to Week 8 or who had all 4 Mayo subscores missing at Week 8 had their last available individual Mayo subscores carried forward. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Baseline and Week 8
Population: PEAS consisted of all participants randomized in the induction study. Here, N (number of participants analyzed) signifies those participants who were analyzed for this OM.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 321
Units on a scale | -1.8 (2.40) | -3.2 (2.81) | -3.5 (2.67)

19. Secondary Outcome: Induction Study - Change From Baseline in Partial Mayo Score Through Week 8
Description: The partial Mayo score, which is sum of 3 subscores of the Mayo score without the endoscopy subscore (stool frequency, rectal bleeding, and physician's global assessment subscores; rated as 0 [normal] to 3 [severe]). The partial Mayo score is calculated as the sum of the 3 subscores and values range from 0 to 9; higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 had their baseline value carried forward from the time of the event onward. Participants with the partial Mayo score missing at a timepoint had their last available individual partial Mayo subscore carried forward to that timepoint.
Time Frame: Baseline through Week 8
Population: PEAS consisted of all participants randomized in the induction study. Here, N (number of participants analyzed) signifies those participants who were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 321
Units on a scale
  Change at Week 2 | -1.0 (1.63) | -1.5 (1.74) | -1.6 (1.69)
  Change at Week 4 | -1.4 (1.86) | -2.1 (1.86) | -2.5 (1.93)
  Change at Week 8 | -1.5 (2.07) | -2.6 (2.31) | -2.9 (2.20)

20. Secondary Outcome: Induction Study - Number of Participants With Individual Mayo Subscore (Stool Frequency) up to Week 8
Description: The stool frequency subscore of Mayo score is rated as 0 (normal) to 3 (severe). Stool frequency scores: 0 =normal number of stools, 1 = 1-2 stools more than normal, 2 = 3-4 stools more than normal, 3 = 5 or more stools more than normal. Higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 had their baseline value carried forward from the time of the event onward. Participants who had a missing Mayo stool frequency subscore at the designated analysis timepoint had the last available value for that subscore carried forward.
Time Frame: Up to Week 8
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 321
Participants
  Week 2:Normal number of stools | 16 | 32 | 26
  Week 2:1-2 stools more than normal | 82 | 99 | 94
  Week 2: 3-4 stools more than normal | 85 | 88 | 90
  Week 2: 5 or more stools more than normal | 136 | 101 | 111
  Week 4:Normal number of stools | 30 | 36 | 50
  Week 4:1-2 stools more than normal | 85 | 122 | 126
  Week 4: 3-4 stools more than normal | 81 | 78 | 72
  Week 4: 5 or more stools more than normal | 123 | 84 | 73
  Week 8:Normal number of stools | 28 | 66 | 71
  Week 8:1-2 stools more than normal | 93 | 112 | 110
  Week 8: 3-4 stools more than normal | 76 | 61 | 85
  Week 8: 5 or more stools more than normal | 122 | 81 | 55

21. Secondary Outcome: Induction Study - Number of Participants With Individual Mayo Subscore (Rectal Bleeding) up to Week 8
Description: The rectal bleeding subscore of the Mayo Score is rated as 0 (normal) to 3 (severe). Rectal bleeding scores: 0 = no blood seen, 1 = streaks of blood with stool less than half the time, 2 = obvious blood with stool most of the time, and 3 = blood alone passed. Higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 had their baseline value carried forward from the time of the event onward. Participants who had a missing Mayo rectal bleeding subscore at the designated analysis timepoint had the last available value for that subscore carried forward.
Time Frame: Up to Week 8
Population: PEAS consisted of all participants randomized in the induction study.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants
  Week 2: No blood seen | 83 | 104 | 120
  Week 2:Streaks of blood with stool < half time | 119 | 122 | 131
  Week 2: Obvious blood with stool most of the time | 94 | 83 | 63
  Week 2: Blood alone passed | 23 | 11 | 8
  Week 4:No blood seen | 117 | 138 | 161
  Week 4:Streaks of blood with stool < half time | 103 | 117 | 115
  Week 4: Obvious blood with stool most of time | 75 | 54 | 40
  Week 4: Blood alone passed | 24 | 11 | 6
  Week 8:No blood seen | 119 | 173 | 204
  Week 8:Streaks of blood with stool < half the time | 106 | 85 | 81
  Week 8: Obvious blood with stool most of the time | 73 | 54 | 31
  Week 8: Blood alone passed | 21 | 8 | 6

22. Secondary Outcome: Induction Study - Number of Participants With Individual Mayo Subscore (Endoscopy Findings) at Week 8
Description: The endoscopy findings subscore of the Mayo score is rated as 0 (normal) to 3 (severe). Endoscopy finding scores: 0 = normal or inactive disease, 1 = mild disease (erythema, decreased vascular pattern, mild friability), 2 = moderate disease (marked erythema, absent vascular pattern, friability, erosions), and 3 = Severe disease (spontaneous bleeding, ulceration). Higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 had their baseline value carried forward from the time of the event onward. Participants who had a missing Mayo endoscopy subscore at Week 8 had the last available value for that subscore carried forward. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 8
Population: PEAS consisted of all participants randomized in the induction study.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants
  Week 8: Normal or inactive disease | 12 | 33 | 25
  Week 8:Mild disease | 32 | 51 | 62
  Week 8: Moderate disease | 99 | 96 | 84
  Week 8: Severe disease | 176 | 140 | 151

23. Secondary Outcome: Induction Study - Number of Participants With Individual Mayo Subscore (Physician's Global Assessment) up to Week 8
Description: The physician's global assessment subscore of the Mayo score is rated as 0 (normal) to 3 (severe). Physician's global assessment scores: 0 = normal, 1 = mild disease, 2 = moderate disease, and 3 = severe disease. Higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 had their baseline value carried forward from the time of the event onward. Participants who had a missing Mayo physician's global assessment subscore at the designated analysis timepoint had the last available value for that subscore carried forward.
Time Frame: Up to Week 8
Population: PEAS consisted of all participants randomized in the induction study.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants
  Week 2: Normal | 3 | 4 | 10
  Week 2:Mild disease | 66 | 82 | 81
  Week 2: Moderate disease | 194 | 193 | 181
  Week 2: Severe disease | 56 | 41 | 50
  Week 4:Normal | 13 | 14 | 22
  Week 4:Mild disease | 82 | 118 | 137
  Week 4: Moderate disease | 181 | 164 | 138
  Week 4: Severe disease | 43 | 24 | 25
  Week 8:Normal | 21 | 37 | 49
  Week 8:Mild disease | 83 | 136 | 135
  Week 8: Moderate disease | 153 | 115 | 106
  Week 8: Severe disease | 62 | 32 | 32

24. Secondary Outcome: Induction Study - Number of Participants With Clinical Remission at Week 8 by Biologic Failure (BF) Status (As Per Global Definition)
Description: Global definition of clinical remission: Mayo score<=2 points, with no individual subscore >1. Mayo score included 4 subscores (stool frequency, rectal bleeding, endoscopy findings, physician's global assessment), rated as 0 (normal) to 3 (severe). Total score = sum of 4 subscores and range from 0 to 12, where 3 to 5 = mild; 6 to 10 = moderate; 11 to 12 = severe; higher scores indicate worsening of disease. BF: participants received treatment with 1 or more tumor necrosis factor (TNF) antagonists and/or vedolizumab at dose approved for treatment of UC and did not respond initially or responded initially but lost response or were intolerant of medication. Participants with prohibited change in concomitant UC medication/ ostomy/colectomy before Week 8 or who had all 4 Mayo subscores missing at Week 8 considered not in clinical remission. Endoscopy subscore assessed during central review of video of endoscopy was used.
Time Frame: Week 8
Population: The primary efficacy analysis set consisted of all participants randomized in the induction study. Here, n (number of participants analyzed) signifies participants analyzed for this OM with specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants
  Participants with BF: number analyzed (Participants) | 161 | 164 | 166
  Participants with BF | 2 | 19 | 21
  Participants without BF: number analyzed (Participants) | 158 | 156 | 156
  Participants without BF | 15 | 31 | 29

25. Secondary Outcome: Induction Study - Number of Participants With Clinical Remission at Week 8 by Biologic Failure (BF) Status (As Per US Definition)
Description: US definition of clinical remission: absolute stool number <=3, a Mayo rectal bleeding subscore of 0 (no blood seen), Mayo endoscopy subscore of (normal/ inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]), without PGA. Absolute stool number: average of daily stool number over 3 days. Mayo rectal bleeding and endoscopy subscores rated 0 (normal) to 3 (severe). BF: participants received treatment with 1/ more TNF antagonists/ vedolizumab at dose approved for treatment of UC, and did not respond initially or responded initially but lost response/ intolerant of medication. Participants with prohibited change in concomitant UC medication/ ostomy/ colectomy before Week 8/ missing all 3 of Mayo components (absolute stool number, rectal bleeding, Mayo endoscopy subscore) at Week 8 considered not in clinical remission. Endoscopy subscore assessed during central review used endoscopy video.
Time Frame: Week 8
Population: PEAS consisted of all participants randomized in the induction study. Here, n (number of participants analyzed) signifies participants analyzed for this OM with specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants
  Participants with BF: number analyzed (Participants) | 161 | 164 | 166
  Participants with BF | 4 | 19 | 22
  Participants without BF: number analyzed (Participants) | 158 | 156 | 156
  Participants without BF | 16 | 34 | 39

26. Secondary Outcome: Induction Study - Number of Participants With Endoscopic Healing at Week 8 by Biologic Failure Status
Description: Number of participants with endoscopic healing at week 8 by BF status were reported. Endoscopic healing is improvement in the endoscopic appearance of the mucosa. It is defined as Mayo endoscopic subscore = 0 (normal or inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]). BF: Participants received treatment with 1/ more TNF antagonists and/or vedolizumab at dose approved for treatment of UC, and either did not respond initially, responded initially but then lost response/ were intolerant of medication. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to Week 8 or who had a missing endoscopy score at Week 8 were considered not to have endoscopic healing. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 8
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants
  Participants with BF: number analyzed (Participants) | 161 | 164 | 166
  Participants with BF | 11 | 30 | 35
  Participants without BF: number analyzed (Participants) | 158 | 156 | 156
  Participants without BF | 33 | 54 | 52

27. Secondary Outcome: Induction Study - Number of Participants With Clinical Response at Week 8 by Biologic Failure Status
Description: Clinical response: decrease from induction baseline in Mayo score by >=30% and >= 3 points, with either decrease from baseline in rectal bleeding subscore >=1/ rectal bleeding subscore= 0/1. Mayo score included 4 subscores (stool frequency, rectal bleeding, endoscopy findings, physician's global assessment), rated as 0 (normal) to 3 (severe). Total score =sum of 4 subscores and range from 0 to 12, where 3 to 5 = mild; 6 to 10 = moderate; 11 to 12 = severe; higher scores =worsening of disease. BF: participants received treatment with 1/ more TNF antagonists and/or vedolizumab at dose approved for treatment of UC, and did not respond initially or responded initially but lost response/ were intolerant of medication. Participants with prohibited change in concomitant UC medication/ ostomy/ colectomy before Week 8 or who had all 4 Mayo subscores missing at Week 8 were considered not in clinical response. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 8
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants
  Participants with BF: number analyzed (Participants) | 161 | 164 | 166
  Participants with BF | 44 | 74 | 95
  Participants without BF: number analyzed (Participants) | 158 | 156 | 156
  Participants without BF | 56 | 90 | 104

28. Secondary Outcome: Induction Study: Number of Participants in Remission Based on Stool Frequency Subscore of 0 or 1, Rectal Bleeding Subscore of 0, and Endoscopy Subscore of 0 or 1 at Week 8 (US Specific)
Description: Number of participants in remission based on stool frequency subscore of 0 (normal number of stools) or 1 (1-2 stools more than normal), rectal bleeding subscore of 0 (no blood seen), and endoscopy subscore of 0 (normal or inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]) at Week 8 were reported. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 or who were missing all 3 of the Mayo components related to this OM (stool frequency, rectal bleeding subscore, and Mayo endoscopy subscore) at Week 8 were considered not to be in remission. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 8
Population: PEAS consisted of all participants randomized in the induction study.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants | 25 | 60 | 67

29. Secondary Outcome: Induction Study: Number of Participants in Remission Based on Stool Frequency Subscore of 0, Rectal Bleeding Subscore of 0, and Endoscopy Subscore of 0 or 1 at Week 8 (US Specific)
Description: Number of participants in remission based on stool frequency subscore of 0 (normal number of stools), rectal bleeding subscore of 0 (no blood seen), and endoscopy subscore of 0 (normal or inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]) at Week 8 were reported. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 or who were missing all 3 of the Mayo components related to this OM (stool frequency, rectal bleeding subscore, and Mayo endoscopy subscore) at Week 8 were considered not to be in remission. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 8
Population: PEAS consisted of all participants randomized in the induction study.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants | 10 | 35 | 29

30. Secondary Outcome: Induction Study - Change From Baseline in C-reactive Protein (CRP) Concentration Through Week 8
Description: Change from baseline in CRP concentration through Week 8 was reported. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to Week 8 had their baseline value carried forward from the time of the event onward. Participants who had a missing CRP value at the designated analysis timepoint had their last value carried forward.
Time Frame: Baseline through Week 8
Population: PEAS consisted of all participants randomized in the induction study. Here, N (number of participants analyzed) signifies participants who were analyzed for this OM.
Measure: Median (Inter-Quartile Range); unit: milligram per liter (mg/L)
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 316 | 315 | 320
milligram per liter (mg/L)
  Change at Week 2 | -0.01 [-2.79 to 1.21] | -0.75 [-4.53 to 0.00] | -0.92 [-6.24 to 0.05]
  Change at Week 4 | -0.18 [-3.12 to 0.71] | -1.08 [-5.86 to 0.00] | -1.94 [-7.16 to -0.06]
  Change at Week 8 | 0.00 [-2.47 to 2.61] | -1.30 [-5.04 to 0.30] | -1.43 [-7.63 to 0.00]

31. Secondary Outcome: Induction Study - Number of Participants With Normalized CRP (<=3 mg/L) up to Week 8 Among Participants With Abnormal CRP (>3 mg/L) at Baseline
Description: Number of participants with normalized CRP (<=3 mg/L) up to Week 8 among participants with abnormal CRP (>3 mg/L) at baseline were reported. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 or who had a missing CRP value at the designated analysis timepoint were considered not to have normalized CRP.
Time Frame: Up to Week 8
Population: PEAS consisted of all participants randomized in the induction study, with those participants who were having abnormal CRP at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 185 | 185 | 199
Participants
  Week 2 | 36 | 54 | 58
  Week 4 | 41 | 70 | 75
  Week 8 | 39 | 63 | 77

32. Secondary Outcome: Induction Study - Change From Baseline in Fecal Lactoferrin Concentration Through Week 8
Description: Change from baseline in fecal lactoferrin concentration through Week 8 was reported. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to Week 8 had their baseline value carried forward from the time of the event onward. Participants who had a missing fecal lactoferrin value at the designated analysis timepoint had their last value carried forward.
Time Frame: Baseline through Week 8
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: microgram per gram (mcg/g)
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 294 | 302 | 306
microgram per gram (mcg/g)
  Change at Week 2 | 0.00 [-103.22 to 120.67] | -4.67 [-140.04 to 75.46] | -24.06 [-202.88 to 60.23]
  Change at Week 4 | 0.00 [-117.67 to 133.67] | -29.26 [-203.79 to 46.29] | -69.51 [-240.62 to 24.90]
  Change at Week 8 | -4.71 [-149.28 to 92.90] | -43.41 [-220.99 to 29.10] | -101.46 [-301.23 to 0.00]

33. Secondary Outcome: Induction Study - Number of Participants With Normalized Fecal Lactoferrin (<=7.24 mcg/g) up to Week 8 Among Participants With Abnormal Fecal Lactoferrin (>7.24 mcg/g) at Baseline
Description: Number of participants with normalized fecal lactoferrin (<=7.24 mcg/g) up to Week 8 among participants with abnormal fecal lactoferrin (> 7.24 mcg/g) at baseline were reported. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 or who had a missing fecal lactoferrin value at the designated analysis timepoint were considered not to have normalized fecal lactoferrin.
Time Frame: Up to Week 8
Population: PEAS consisted of all participants randomized in the induction study, with those participants who had abnormal fecal lactoferrin at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 280 | 291 | 294
Participants
  Week 2 | 16 | 17 | 15
  Week 4 | 16 | 37 | 33
  Week 8 | 26 | 50 | 43

34. Secondary Outcome: Induction Study - Change From Baseline in Fecal Calprotectin Concentration Through Week 8
Description: Change from baseline in fecal calprotectin concentration through Week 8 was reported. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to Week 8 had their baseline value carried forward from the time of the event onward. Participants who had a missing fecal calprotectin value at the designated analysis timepoint had their last value carried forward.
Time Frame: Baseline through Week 8
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: milligram per kilogram (mg/kg)
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 289 | 296 | 300
milligram per kilogram (mg/kg)
  Change at Week 2 | 0.00 [-702.00 to 631.00] | -29.00 [-933.50 to 492.00] | -127.00 [-1029.50 to 433.50]
  Change at Week 4 | -2.00 [-961.00 to 894.00] | -223.00 [-1200.50 to 266.50] | -485.50 [-1536.50 to 158.50]
  Change at Week 8 | -59.00 [-996.00 to 751.00] | -431.50 [-1635.50 to 175.00] | -715.50 [-1913.50 to 0.00]

35. Secondary Outcome: Induction Study - Number of Participants With Normalized Fecal Calprotectin (<=250 mg/kg) up to Week 8 Among Participants With Abnormal Fecal Calprotectin (>250 mg/kg) at Baseline
Description: Number of participants with normalized fecal calprotectin (<=250 milligram per kilogram [mg/kg) up to Week 8 among participants with abnormal fecal calprotectin (>250 mg/kg) at baseline were reported. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 or who had a missing fecal calprotectin value at the designated analysis timepoint were considered not to have normalized fecal calprotectin.
Time Frame: Up to Week 8
Population: PEAS consisted of all randomized participants in the induction study, with abnormal fecal calprotectin (>250 mg/kg) at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 250 | 264 | 274
Participants
  Week 2 | 20 | 37 | 37
  Week 4 | 25 | 45 | 47
  Week 8 | 51 | 64 | 70

36. Secondary Outcome: Induction Study - Number of Participants With a >20-point Improvement From Baseline in Total Inflammatory Bowel Disease Questionnaire (IBDQ) Score at Week 8
Description: The IBDQ is 32-item questionnaire for participants with Inflammatory Bowel Disease (IBD) used to evaluate disease-specific health-related quality of life. IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). The 32 items were grouped into 4 domains: bowel function, emotional status, systemic symptoms and social function. The 4 domains were scored as follows: 10 to 70 (bowel symptoms); 5 to 35 (systemic symptoms); 12 to 84 (emotional function); and 5 to 35 (social function). For each domain, higher score indicated better quality of life. Total score is sum of each item score and ranges from 32 to 224 with higher score indicating better quality of life. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy prior to the Week 8 or who had a missing IBDQ score at either baseline or Week 8 were considered not to have achieved a greater than 20-point improvement.
Time Frame: Baseline and Week 8
Population: PEAS consisted of all participants randomized in the induction study.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Participants | 118 | 196 | 200

37. Secondary Outcome: Induction Study - Change From Baseline in IBDQ Dimension Scores at Week 8
Description: The IBDQ is 32-item questionnaire for participants with IBD used to evaluate disease-specific health-related quality of life. IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). The 32 items were grouped into 4 domains: bowel function, emotional status, systemic symptoms and social function. The 4 domains were scored as: 10 to 70 (bowel symptoms); 5 to 35 (systemic symptoms); 12 to 84 (emotional function); and 5 to 35 (social function). For each domain, higher score indicated better quality of life. Total score is sum of each item score and ranges from 32 to 224 with higher score indicating better quality of life. Participants who had prohibited change in concomitant UC medication or ostomy or colectomy prior to Week 8 had their baseline value carried forward from time of event onward and participants who had missing IBDQ dimension score at designated analysis timepoint had their last value carried forward.
Time Frame: Baseline and Week 8
Population: PEAS consisted of all participants randomized in the induction study. Here, n (number of participants analyzed) signifies participants who were analyzed for this OM at specified category.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Units on a scale
  Bowel: Change at Week 8: number analyzed (Participants) | 317 | 319 | 321
  Bowel: Change at Week 8 | 5.9 (10.34) | 12.5 (11.27) | 12.7 (11.11)
  Emotional: Change at Week 8: number analyzed (Participants) | 317 | 317 | 321
  Emotional: Change at Week 8 | 5.3 (12.33) | 10.1 (12.39) | 11.2 (12.33)
  Systemic: Change at Week 8: number analyzed (Participants) | 317 | 319 | 321
  Systemic: Change at Week 8 | 2.3 (5.59) | 5.1 (5.59) | 5.2 (5.65)
  Social: Change at Week 8: number analyzed (Participants) | 317 | 318 | 321
  Social: Change at Week 8 | 2.7 (6.55) | 5.7 (7.41) | 5.9 (6.44)

38. Secondary Outcome: Induction Study - Change From Baseline in 36-Item Short-Form (SF-36) Physical Component Score (PCS) and Mental Component Score (MCS) at Week 8
Description: SF-36 evaluates 8 individual subscales (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health). Each 8 scales scored from 0 to 100 with higher scores= better health. Based on scale scores, physical component summary (PCS: calculated from subscales physical functioning, role-physical, bodily pain, and general health) and mental component summary (MCS: calculated from subscales vitality, social functioning, role-emotional and mental health) scores were derived. Summary MCS and PCS score is also scaled from 0 to 100 with higher scores= better health. Participants who had prohibited change in concomitant UC medication or an ostomy or colectomy prior to Week 8 had their baseline value carried forward from time of event onward or participants who had missing component summary score at Week 8 had their last value carried forward.
Time Frame: Baseline and Week 8
Population: PEAS consisted of all participants randomized in the induction study. Here, n (number of participants analyzed) signifies participants who were analyzed for this OM at specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Units on a scale
  PCS: Change at Week 8: number analyzed (Participants) | 319 | 318 | 322
  PCS: Change at Week 8 | 2.1 (6.39) | 4.7 (6.49) | 5.2 (6.16)
  MCS: Change at Week 8: number analyzed (Participants) | 319 | 318 | 322
  MCS: Change at Week 8 | 2.2 (10.20) | 5.3 (9.63) | 5.1 (9.72)

39. Secondary Outcome: Induction Study - Change From Baseline in Individual Subscales of 36-Item Short-Form (SF-36) at Week 8
Description: SF-36 evaluates 8 individual subscales (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health). Each 8 scales scored from 0 to 100 with higher scores= better health. Participants who had prohibited change in concomitant UC medication or an ostomy or colectomy prior to Week 8 had their baseline value carried forward from time of event onward or participants who had missing individual scale at a designated analysis timepoint had their last value carried forward.
Time Frame: Baseline and Week 8
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 318 | 322
Units on a scale
  Physical functioning: Change at Week 8 | 1.7 (6.46) | 3.0 (6.46) | 3.4 (6.51)
  Role-physical: Change at Week 8 | 2.4 (9.51) | 5.9 (9.34) | 6.1 (8.53)
  Bodily pain: Change at Week 8 | 2.6 (9.71) | 6.0 (9.45) | 6.8 (9.08)
  General health: Change at Week 8 | 1.5 (7.36) | 4.7 (7.74) | 4.5 (7.10)
  Vitality: Change at Week 8 | 2.7 (9.93) | 6.1 (9.35) | 6.8 (9.78)
  Social functioning: Change at Week 8 | 3.0 (10.52) | 6.6 (10.25) | 6.4 (9.84)
  Role-emotional: Change at Week 8 | 1.6 (11.04) | 4.4 (11.04) | 3.6 (10.53)
  Mental health: Change at Week 8 | 2.0 (9.86) | 4.7 (9.14) | 5.1 (9.27)

40. Secondary Outcome: Induction Study - Change From Baseline in EuroQOL-5 Dimensions (EQ-5D) Health Questionnaire Index Score at Week 8
Description: EQ-5D descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). The responses to 5 EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 (death) to 1 (full health). Participants who had prohibited change in concomitant UC medication or an ostomy or colectomy prior to Week 8 had their baseline value carried forward from time of event onward or participants who had missing score at a designated analysis timepoint had their last value carried forward.
Time Frame: Baseline and Week 8
Population: PEAS consisted of all participants randomized in the induction study. Here, N (number of participants analyzed) signifies participants analyzed for this OM.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 317 | 319 | 322
Units on a scale | 0.04 (0.182) | 0.09 (0.182) | 0.11 (0.172)

41. Secondary Outcome: Induction Study - Change From Baseline in EuroQOL-5 Dimensions (EQ-5D) Health State Visual Analog Scale (VAS) Score at Week 8
Description: The EQ-5D VAS records the participant's self-rated health on a vertical, VAS, with 0 representing the worst imaginable health state and 100 representing the best imaginable health state. The EQ VAS is used as a quantitative measure of health outcome as judged by the individual participant. Participants who had prohibited change in concomitant UC medication or an ostomy or colectomy prior to Week 8 had their baseline value carried forward from time of event onward or participants who had missing score at a designated analysis timepoint had their last value carried forward.
Time Frame: Baseline and Week 8
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 317 | 319 | 322
Units on a scale | 5.71 (19.584) | 13.64 (20.394) | 13.51 (18.447)

42. Secondary Outcome: Induction Study - Percentage of Participants With Change From Baseline in EuroQOL-5 Dimensions (EQ-5D) Score at Week 8
Description: EQ-5D descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). The responses to 5 EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 (death) to 1 (full health). Participants who had prohibited change in concomitant UC medication or an ostomy or colectomy prior to Week 8 had their baseline value carried forward from time of event onward or participants who had missing score at a designated analysis timepoint had their last value carried forward. Percentage of participants with various responses to the 5 dimensions were reported.
Time Frame: Baseline and Week 8
Population: as for outcome 37
Measure: Number; unit: Percentage of Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6 mg/kg IV
Number analyzed (Participants) | 319 | 320 | 322
Percentage of Participants
  Mobility:Improved at Week 8: number analyzed (Participants) | 317 | 319 | 322
  Mobility:Improved at Week 8 | 18.0 | 16.3 | 24.2
  Mobility:No change at Week 8: number analyzed (Participants) | 317 | 319 | 322
  Mobility:No change at Week 8 | 71.9 | 71.8 | 66.8
  Mobility:Worsened at Week 8: number analyzed (Participants) | 317 | 319 | 322
  Mobility:Worsened at Week 8 | 10.1 | 11.9 | 9.0
  Self-care:Improved at Week 8: number analyzed (Participants) | 317 | 319 | 322
  Self-care:Improved at Week 8 | 5.4 | 6.9 | 7.5
  Self-care:No change at Week 8: number analyzed (Participants) | 317 | 319 | 322
  Self-care:No change at Week 8 | 89.6 | 88.4 | 90.4
  Self-care:Worsened at Week 8: number analyzed (Participants) | 317 | 319 | 322
  Self-care:Worsened at Week 8 | 5.0 | 4.7 | 2.2
  Usual activities:Improved at Week 8: number analyzed (Participants) | 317 | 319 | 322
  Usual activities:Improved at Week 8 | 34.1 | 49.5 | 45.0
  Usual activities:No Change at Week 8: number analyzed (Participants) | 317 | 319 | 322
  Usual activities:No Change at Week 8 | 51.1 | 40.4 | 44.1
  Usual activities:Worsened at Week 8: number analyzed (Participants) | 317 | 319 | 322
  Usual activities:Worsened at Week 8 | 14.8 | 10.0 | 10.9
  Pain/discomfort: Improved at Week 8 | 34.4 | 44.2 | 43.5
  Pain/discomfort: No Change at Week 8: number analyzed (Participants) | 317 | 319 | 322
  Pain/discomfort: No Change at Week 8 | 49.8 | 48.3 | 48.1
  Pain/discomfort: Worsened at Week 8: number analyzed (Participants) | 317 | 319 | 322
  Pain/discomfort: Worsened at Week 8 | 15.8 | 7.5 | 8.4
  Anxiety/depression: Improved at Week 8: number analyzed (Participants) | 317 | 319 | 322
  Anxiety/depression: Improved at Week 8 | 26.8 | 33.5 | 37.6
  Anxiety/depression: No Change at Week 8: number analyzed (Participants) | 317 | 319 | 322
  Anxiety/depression: No Change at Week 8 | 55.5 | 54.2 | 51.6
  Anxiety/depression: Worsened at Week 8: number analyzed (Participants) | 317 | 319 | 322
  Anxiety/depression: Worsened at Week 8 | 17.7 | 12.2 | 10.9

43. Secondary Outcome: Maintenance Study - Change From Maintenance Baseline in Mayo Score at Week 44
Description: The Mayo score consists of 4 subscores (stool frequency, rectal bleeding, endoscopy findings, and physician's global assessment), rated as 0 (normal) to 3 (severe). Total score is calculated as the sum of 4 subscores and values range from 0 to 12 scores, where 3 to 5 = mild; 6 to 10 = moderate; and 11 to 12 = severe; higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy , or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to Week 44 had their Week 0 value of the induction study carried forward or who had all 4 Mayo subscores missing at Week 44 had their last available individual Mayo subscores carried forward. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Baseline and Week 44
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Units on a scale | 1.6 (3.45) | 0.1 (3.02) | -0.5 (2.88)

44. Secondary Outcome: Maintenance Study - Change From Induction Baseline in Mayo Score at Week 44
Description: The Mayo score consists of 4 subscores (stool frequency, rectal bleeding, endoscopy findings, and physician's global assessment), rated as 0 (normal) to 3 (severe). Total Mayo score is calculated as the sum of 4 subscores and values range from 0 to 12 scores, where 3 to 5 = mild; 6 to 10 = moderate; and 11 to 12 = severe; higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 had their Week 0 value of the induction study carried forward from the time of the event onward or who had all 4 Mayo subscores missing at Week 44 had their last available individual Mayo subscores carried forward. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Induction Baseline and Week 44
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Units on a scale | -3.3 (3.34) | -5.0 (3.27) | -5.6 (3.17)

45. Secondary Outcome: Maintenance Study - Number of Participants With Individual Mayo Subscore (Stool Frequency) up to Week 44
Description: Stool frequency subscore of Mayo score is rated as 0 (normal) to 3 (severe). Stool frequency scores: 0 =normal number of stools, 1 = 1-2 stools more than normal, 2 = 3-4 stools more than normal, 3 = 5 or more stools more than normal. Higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 had their Week 0 value of the induction study carried forward from the time of the event onward or who had a missing Mayo subscores at a timepoint had the last available value for that subscore carried forward.
Time Frame: Up to Week 44
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants
  Week 4:Normal number of stools | 56 | 61 | 58
  Week 4:1-2 stools more than normal | 91 | 76 | 86
  Week 4: 3-4 stools more than normal | 21 | 26 | 29
  Week 4: 5 or more stools more than normal | 7 | 9 | 3
  Week 8:Normal number of stools | 70 | 62 | 61
  Week 8:1-2 stools more than normal | 69 | 75 | 84
  Week 8: 3-4 stools more than normal | 22 | 25 | 26
  Week 8: 5 or more stools more than normal | 14 | 10 | 5
  Week 12:Normal number of stools | 62 | 55 | 64
  Week 12:1-2 stools more than normal | 72 | 75 | 85
  Week 12: 3-4 stools more than normal | 20 | 28 | 21
  Week 12: 5 or more stools more than normal | 21 | 14 | 6
  Week 16:Normal number of stools | 63 | 51 | 73
  Week 16:1-2 stools more than normal | 66 | 78 | 77
  Week 16: 3-4 stools more than normal | 25 | 27 | 15
  Week 16: 5 or more stools more than normal | 21 | 16 | 11
  Week 20:Normal number of stools | 59 | 63 | 67
  Week 20:1-2 stools more than normal | 55 | 65 | 85
  Week 20: 3-4 stools more than normal | 34 | 26 | 15
  Week 20: 5 or more stools more than normal | 27 | 18 | 9
  Week 24:Normal number of stools | 50 | 64 | 72
  Week 24:1-2 stools more than normal | 63 | 61 | 73
  Week 24: 3-4 stools more than normal | 31 | 31 | 20
  Week 24: 5 or more stools more than normal | 31 | 16 | 11
  Week 28:Normal number of stools | 52 | 64 | 67
  Week 28:1-2 stools more than normal | 53 | 64 | 76
  Week 28: 3-4 stools more than normal | 34 | 24 | 22
  Week 28: 5 or more stools more than normal | 36 | 20 | 11
  Week 32:Normal number of stools | 51 | 59 | 72
  Week 32:1-2 stools more than normal | 55 | 66 | 73
  Week 32: 3-4 stools more than normal | 35 | 25 | 18
  Week 32: 5 or more stools more than normal | 34 | 22 | 13
  Week 36:Normal number of stools | 49 | 59 | 77
  Week 36:1-2 stools more than normal | 52 | 60 | 66
  Week 36: 3-4 stools more than normal | 36 | 29 | 18
  Week 36: 5 or more stools more than normal | 38 | 24 | 15
  Week 40:Normal number of stools | 49 | 55 | 81
  Week 40:1-2 stools more than normal | 50 | 65 | 58
  Week 40: 3-4 stools more than normal | 36 | 26 | 21
  Week 40: 5 or more stools more than normal | 40 | 26 | 16
  Week 44:Normal number of stools | 46 | 62 | 71
  Week 44:1-2 stools more than normal | 53 | 57 | 72
  Week 44: 3-4 stools more than normal | 35 | 28 | 16
  Week 44: 5 or more stools more than normal | 41 | 25 | 17

46. Secondary Outcome: Maintenance Study - Number of Participants With Individual Mayo Subscore (Rectal Bleeding) up to Week 44
Description: The rectal bleeding subscore of the Mayo Score is rated as 0 (normal) to 3 (severe). Rectal bleeding scores: 0 = no blood seen, 1 = streaks of blood with stool <half time, 2 = obvious blood with stool most of time, and 3 = blood alone passed. Higher scores = worsening of disease. Participants who had prohibited change in concomitant UC medication/ ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study agent due to lack of therapeutic effect/ due to AE of worsening of UC before Week 44 had their Week 0 value of induction study carried forward from time of event onward and who had missing Mayo subscores at timepoint had last available value for that subscore carried forward.
Time Frame: Up to Week 44
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants
  Week 4:No blood seen | 149 | 148 | 143
  Week 4:Streaks of blood with stool < half time | 20 | 23 | 29
  Week 4: Obvious blood with stool most of the time | 4 | 1 | 24
  Week 4: Blood alone passed | 2 | 0 | 0
  Week 8:No blood seen | 139 | 151 | 141
  Week 8:Streaks of blood with stool < half time | 27 | 17 | 31
  Week 8: Obvious blood with stool most of time | 6 | 3 | 4
  Week 8:Blood alone passed | 3 | 1 | 0
  Week 12:No blood seen | 141 | 144 | 149
  Week 12:Streaks of blood with stool <half time | 21 | 19 | 18
  Week 12: Obvious blood with stool most of the time | 10 | 8 | 6
  Week 12: Blood alone passed | 3 | 1 | 3
  Week 16:No blood seen | 134 | 145 | 150
  Week 16:Streaks of blood with stool < half time | 24 | 17 | 17
  Week 16: Obvious blood with stool most of the time | 13 | 8 | 8
  Week 16: Blood alone passed | 4 | 2 | 1
  Week 20:No blood seen | 120 | 141 | 144
  Week 20:Streaks of blood with stool <half time | 31 | 17 | 20
  Week 20: Obvious blood with stool most of the time | 19 | 12 | 11
  Week 20: Blood alone passed | 5 | 2 | 1
  Week 24:No blood seen | 114 | 139 | 144
  Week 24:Streaks of blood with stool <half time | 32 | 18 | 19
  Week 24: Obvious blood with stool most of the time | 23 | 12 | 11
  Week 24: Blood alone passed | 6 | 3 | 2
  Week 28:No blood seen | 114 | 141 | 147
  Week 28:Streaks of blood with stool <half time | 26 | 18 | 12
  Week 28: Obvious blood with stool most of the time | 28 | 10 | 14
  Week 28: Blood alone passed | 7 | 3 | 3
  Week 32:No blood seen | 109 | 138 | 147
  Week 32:Streaks of blood with stool <half time | 32 | 16 | 13
  Week 32: Obvious blood with stool most of the time | 25 | 14 | 14
  Week 32: Blood alone passed | 9 | 4 | 2
  Week 36:No blood seen | 108 | 136 | 150
  Week 36:Streaks of blood with stool <half time | 30 | 18 | 9
  Week 36: Obvious blood with stool most of the time | 28 | 15 | 15
  Week 36: Blood alone passed | 9 | 3 | 2
  Week 40:No blood seen | 105 | 132 | 147
  Week 40:Streaks of blood with stool <half time | 33 | 22 | 10
  Week 40: Obvious blood with stool most of the time | 28 | 13 | 17
  Week 40: Blood alone passed | 9 | 5 | 2
  Week 44:No blood seen | 101 | 137 | 139
  Week 44::Streaks of blood with stool <half time | 35 | 15 | 16
  Week 44: Obvious blood with stool most of the time | 30 | 15 | 19
  Week 44: Blood alone passed | 9 | 5 | 2

47. Secondary Outcome: Maintenance Study - Number of Participants With Individual Mayo Subscore (Endoscopy Findings) at Week 44
Description: The endoscopy findings subscore of the Mayo score is rated as 0 (normal) to 3 (severe). Endoscopy finding scores: 0 =normal/ inactive disease, 1 =mild disease (erythema, decreased vascular pattern, mild friability), 2 =moderate disease (marked erythema, absent vascular pattern, friability, erosions), and 3 =severe disease (spontaneous bleeding, ulceration). Higher scores = worsening of disease. Participants who had prohibited change in concomitant UC medication/ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study agent due to lack of therapeutic effect/ AE of worsening of UC before Week 44 had Week 0 value of induction study carried forward from time of event onward and who had missing endoscopy subscores at timepoint had last available value for that subscore carried forward. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 44
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants
  Week 44: Normal or inactive disease | 33 | 43 | 52
  Week 44:Mild disease | 21 | 37 | 42
  Week 44: Moderate disease | 40 | 42 | 50
  Week 44: Severe disease | 81 | 50 | 32

48. Secondary Outcome: Maintenance Study - Number of Participants With Individual Mayo Subscore (Physician's Global Assessment) up to Week 44
Description: The physician's global assessment subscore of the Mayo score is rated as 0 (normal) to 3 (severe). Physician's global assessment scores: 0 = normal, 1 = mild disease, 2 = moderate disease, and 3 = severe disease. Higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 had their Week 0 value of the induction study carried forward from the time of the event onward and who had a missing Mayo subscores at a timepoint had the last available value for that subscore carried forward.
Time Frame: Up to Week 44
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Study (IS): Placebo Intravenous (IV) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants
  Week 4:Normal | 62 | 61 | 59
  Week 4:Mild disease | 100 | 99 | 105
  Week 4: Moderate disease | 12 | 12 | 11
  Week 4: Severe disease | 1 | 0 | 1
  Week 8:Normal | 65 | 70 | 76
  Week 8:Mild disease | 90 | 89 | 88
  Week 8: Moderate disease | 17 | 13 | 11
  Week 8:Severe disease | 3 | 0 | 1
  Week 12:Normal | 66 | 68 | 73
  Week 12:Mild disease | 79 | 81 | 88
  Week 12: Moderate disease | 26 | 16 | 14
  Week 12: Severe disease | 4 | 7 | 1
  Week 16:Normal | 67 | 82 | 83
  Week 16:Mild disease | 68 | 69 | 78
  Week 16: Moderate disease | 32 | 14 | 13
  Week 16: Severe disease | 8 | 7 | 2
  Week 20:Normal | 65 | 85 | 84
  Week 20:Mild disease | 57 | 63 | 73
  Week 20: Moderate disease | 41 | 16 | 16
  Week 20: Severe disease | 12 | 8 | 3
  Week 24:Normal | 54 | 84 | 91
  Week 24:Mild disease | 61 | 65 | 68
  Week 24: Moderate disease | 44 | 14 | 15
  Week 24: Severe disease | 16 | 9 | 2
  Week 28:Normal | 58 | 86 | 89
  Week 28:Mild disease | 52 | 63 | 65
  Week 28: Moderate disease | 47 | 14 | 20
  Week 28: Severe disease | 18 | 9 | 2
  Week 32:Normal | 55 | 84 | 92
  Week 32:Mild disease | 52 | 56 | 62
  Week 32: Moderate disease | 46 | 23 | 19
  Week 32: Severe disease | 22 | 9 | 3
  Week 36: Normal | 59 | 78 | 93
  Week 36:Mild disease | 45 | 60 | 60
  Week 36: Moderate disease | 47 | 24 | 19
  Week 36: Severe disease | 24 | 10 | 4
  Week 40:Normal | 57 | 83 | 91
  Week 40:Mild disease | 48 | 50 | 60
  Week 40: Moderate disease | 44 | 24 | 21
  Week 40: Severe disease | 26 | 15 | 4
  Week 44:Normal | 47 | 78 | 85
  Week 44:Mild disease | 44 | 54 | 62
  Week 44:Moderate disease | 57 | 24 | 25
  Week 44: Severe disease | 27 | 16 | 4

49. Secondary Outcome: Maintenance Study - Change From Maintenance Baseline in Partial Mayo Score Through Week 44
Description: The partial Mayo score, which is sum of 3 subscores of the Mayo score without the endoscopy subscore (stool frequency, rectal bleeding, and physician's global assessment subscores), rated as 0 (normal) to 3 (severe). The partial Mayo score is calculated as the sum of the 3 subscores and values range from 0 to 9; higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 had their Week 0 value of the induction study carried forward from the time of the event onward. Participants who had a missing partial Mayo score at a time point had their last available individual partial Mayo subscore carried forward to that time point.
Time Frame: Baseline through Week 44
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Units on a scale
  Change at Week 4 | -0.2 (1.24) | -0.3 (1.23) | -0.1 (1.26)
  Change at Week 8 | -0.1 (1.59) | -0.3 (1.15) | -0.2 (1.44)
  Change at Week 12 | 0.1 (1.82) | 0.0 (1.66) | -0.2 (1.63)
  Change at Week 16 | 0.3 (2.07) | -0.1 (1.76) | -0.3 (1.76)
  Change at Week 20 | 0.6 (2.36) | -0.1 (1.91) | -0.2 (1.92)
  Change at Week 24 | 0.9 (2.34) | 0.0 (2.02) | -0.3 (1.88)
  Change at Week 28 | 1.0 (2.53) | -0.1 (1.95) | -0.2 (1.94)
  Change at Week 32 | 1.1 (2.60) | 0.1 (2.12) | -0.2 (1.96)
  Change at Week 36 | 1.2 (2.62) | 0.2 (2.13) | -0.2 (2.08)
  Change at Week 40 | 1.3 (2.64) | 0.3 (2.27) | -0.2 (1.97)
  Change at Week 44 | 1.5 (2.63) | 0.3 (2.29) | 0.0 (2.09)

50. Secondary Outcome: Maintenance Study - Change From Induction Baseline in Partial Mayo Score Through Week 44
Description: The partial Mayo score, which is sum of 3 subscores of the Mayo score without the endoscopy subscore (stool frequency, rectal bleeding, and physician's global assessment subscores; rated as 0 [normal] to 3 [severe]). The partial Mayo score is calculated as the sum of the 3 subscores and values range from 0 to 9; higher scores indicate worsening of the disease. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 had their Week 0 value of the induction study carried forward from the time of the event onward. Participants who had a missing partial Mayo score at a time point had their last available individual partial Mayo subscore carried forward to that time point.
Time Frame: Baseline through Week 44
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Units on a scale
  Change at Week 4 | -4.2 (1.70) | -4.5 (1.76) | -4.4 (1.72)
  Change at Week 8 | -4.1 (1.80) | -4.5 (1.68) | -4.5 (1.85)
  Change at Week 12 | -3.9 (2.07) | -4.2 (2.02) | -4.5 (2.02)
  Change at Week 16 | -3.7 (2.17) | -4.3 (2.07) | -4.6 (2.08)
  Change at Week 20 | -3.4 (2.26) | -4.3 (2.13) | -4.5 (2.13)
  Change at Week 24 | -3.1 (2.36) | -4.2 (2.26) | -4.5 (2.18)
  Change at Week 28 | -3.0 (2.49) | -4.3 (2.26) | -4.4 (2.27)
  Change at Week 32 | -2.9 (2.51) | -4.1 (2.40) | -4.5 (2.30)
  Change at Week 36 | -2.8 (2.43) | -4.0 (2.43) | -4.5 (2.40)
  Change at Week 40 | -2.7 (2.51) | -3.9 (2.46) | -4.5 (2.39)
  Change at Week 44 | -2.5 (2.52) | -3.9 (2.49) | -4.3 (2.48)

51. Secondary Outcome: Maintenance Study: Number of Participants in Remission Based on Stool Frequency Subscore of 0 or 1, Rectal Bleeding Subscore of 0, and Endoscopy Subscore of 0 or 1 at Week 44
Description: Number of participants in remission based on stool frequency subscore of 0 (normal number of stools) or 1 (1-2 stools more than normal), rectal bleeding subscore of 0 (no blood seen), and endoscopy subscore of 0 (normal or inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]) at Week 44 were reported. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 and who were missing all 3 of the Mayo subscores related to this OM (stool frequency, rectal bleeding subscore, and Mayo endoscopy subscore) at Week 44 were considered not to be in remission. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 44
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants | 49 | 70 | 84

52. Secondary Outcome: Maintenance Study: Number of Participants in Remission Based on Stool Frequency Subscore of 0, Rectal Bleeding Subscore of 0, and Endoscopy Subscore of 0 or 1 at Week 44
Description: Number of participants in remission based on stool frequency subscore of 0 (normal number of stools), rectal bleeding subscore of 0 (no blood seen), and endoscopy subscore of 0 (normal or inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]) at Week 44 were reported. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 or who were missing all 3 of the Mayo subscores related to this OM (stool frequency, rectal bleeding subscore, and Mayo endoscopy subscore) at Week 44 were considered not to be in remission. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 44
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants | 30 | 42 | 48

53. Secondary Outcome: Maintenance Study: Number of Participants in Symptomatic Remission at Week 44
Description: Symptomatic remission was defined as a Mayo stool frequency subscore of 0 (normal number of stools) or 1 (1-2 stools more than normal) and a rectal bleeding subscore of 0 (no blood seen). Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 were considered not to be in symptomatic remission from the time of the event onward. Participants who had both stool frequency and rectal bleeding subscores missing at Week 44 were considered not to be in symptomatic remission for that visit. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 44
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants | 79 | 107 | 119

54. Secondary Outcome: Maintenance Study: Number of Participants With Clinical Remission at Week 44 by Biologic Failure Status (As Per Global Definition)
Description: Global definition of clinical remission: Mayo score <=2 points, with no individual subscore >1. Mayo score included 4 subscores (stool frequency, rectal bleeding, endoscopy findings, physician's global assessment), rated as 0 (normal) to 3 (severe). Total score =sum of 4 subscores and range from 0 to 12, where 3 to 5=mild; 6 to 10=moderate; 11 to 12=severe; higher scores=worsening of disease. BF: participants received treatment with 1/ more TNF antagonists/ vedolizumab at dose approved for treatment of UC, and did not respond initially or responded initially but lost response/ were intolerant of medication. Participants with prohibited change in UC medication/ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study drug due to lack of therapeutic effect/ AE of worsening of UC before Week 44 or who had all 4 Mayo subscores missing at Week 44 considered not in clinical remission. Endoscopy subscore assessed during central review of video of endoscopy was used.
Time Frame: Week 44
Population: PEAS consisted of all participants who were in clinical response to IV ustekinumab induction and were randomized at Week 0 of the maintenance study to ustekinumab 90 mg SC q8w, ustekinumab 90 mg SC q12w, or placebo SC. Here, n (number of participants analyzed) signifies participants who were analyzed for this OM with specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants
  Participants with BF: number analyzed (Participants) | 88 | 70 | 91
  Participants with BF | 15 | 16 | 36
  Participants without BF: number analyzed (Participants) | 87 | 102 | 85
  Participants without BF | 27 | 50 | 41

55. Secondary Outcome: Maintenance Study: Number of Participants With Clinical Remission at Week 44 by Biologic Failure Status (As Per US Definition)
Description: US definition of clinical remission: absolute stool number <=3, Mayo rectal bleeding subscore: 0 (no blood seen), Mayo endoscopy subscore: 0(normal/ inactive disease) or 1(mild disease [erythema, decreased vascular pattern, mild friability]). Absolute stool number: average of daily stool number over 3 days. Mayo rectal bleeding and endoscopy subscores: 0(normal) to 3(severe). BF: participants received 1/ more TNF antagonists/ vedolizumab for treatment of UC, not responded initially/ responded initially but lost response/ were intolerant of medicines. Participants with prohibited change in UC medication/ ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study drug due to lack of therapeutic effect /due to AE of worsening of UC before Week 44 or who were missing all 3 of Mayo components (absolute stool number, rectal bleeding and endoscopy) at Week 44 were not in clinical remission. Endoscopy subscore assessed during central review used video of endoscopy.
Time Frame: Week 44
Population: as for outcome 54
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants
  Participants with BF: number analyzed (Participants) | 88 | 70 | 91
  Participants with BF | 15 | 17 | 34
  Participants without BF: number analyzed (Participants) | 87 | 102 | 85
  Participants without BF | 28 | 51 | 41

56. Secondary Outcome: Maintenance Study: Number of Participants With Clinical Response up to Week 44 by Biologic Failure Status
Description: Clinical response: decrease from IS baseline in Mayo score by >=30% and >=3 points, with either decrease from baseline in RB subscore >=1/ RB subscore of 0/ 1. Mayo score have 4 subscores (SF, RB, endoscopy findings, PGA), rated 0(normal) to 3(severe). Total score=sum of 4 subscores and range from 0 to 12, where 3 to 5=mild; 6 to 10=moderate; 11 to 12=severe; higher scores=worsening of disease. BF: participants received treatment: 1/ more TNF antagonists/ vedolizumab for treating UC, no respond initially/responded initially but lost response/ medication intolerant. Participants with prohibited change in concomitant UC medication/ ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study drug due to lack of therapeutic effect/ AE of worsen UC before Week 44, had all 4 Mayo subscores miss at Week44/ lost clinical response at any time before Week44 were not in clinical response upto Week44. Endoscopy subscore assessed during central review used endoscopy video.
Time Frame: Up to Week 44
Population: PEAS consisted of all participants who were in clinical response to IV ustekinumab induction and were randomized at Week 0 of the maintenance study to ustekinumab 90 mg SC q8w, ustekinumab 90 mg SC q12w, or placebo SC. Here, n (number of participants analyzed) signifies participants analyzed for this OM with specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants
  Participants with BF: number analyzed (Participants) | 88 | 70 | 91
  Participants with BF | 34 | 39 | 59
  Participants without BF: number analyzed (Participants) | 87 | 102 | 85
  Participants without BF | 44 | 78 | 66

57. Secondary Outcome: Maintenance Study: Number of Participants With Endoscopic Healing at Week 44 by Biologic Failure Status
Description: Number of participants with endoscopic healing at week 44 by BF status were reported. Endoscopic healing is improvement in endoscopic appearance of mucosa. It is defined as Mayo endoscopic subscore = 0 (normal or inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]). BF: participants received treatment with 1 or more tumor necrosis factor (TNF) antagonists or vedolizumab at dose approved for treatment of UC, and either did not respond initially, responded initially but then lost response, or were intolerant of medication. Participants who had prohibited change in concomitant UC medication or ostomy or colectomy, or used rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to AE of worsening of UC prior to Week 44 or who had missing endoscopy score at Week 44 were considered not to have endoscopic healing. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 44
Population: as for outcome 56
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants
  Participants with BF: number analyzed (Participants) | 88 | 70 | 91
  Participants with BF | 20 | 18 | 41
  Participants without BF: number analyzed (Participants) | 87 | 102 | 85
  Participants without BF | 30 | 57 | 49

58. Secondary Outcome: Maintenance Study: Number of Participants With Endoscopic Healing at Week 44 Among Participants Who Had Achieved Endoscopic Healing at Maintenance Baseline
Description: Endoscopic healing is improvement in the endoscopic appearance of the mucosa. It is defined as Mayo endoscopic subscore = 0 (normal or inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]). Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 or who had a missing endoscopy score at Week 44 were considered not to have endoscopic healing. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 44
Population: PEAS consisted of all participants who were in clinical response to IV ustekinumab induction and were randomized at Week 0 of the maintenance study to ustekinumab 90 mg SC q8w, ustekinumab 90 mg SC q12w, or placebo SC, with participants who had achieved endoscopic healing at maintenance baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 71 | 68 | 57
Participants | 25 | 41 | 37

59. Secondary Outcome: Maintenance Study: Number of Participants With Normal or Inactive Mucosal Disease at Week 44
Description: Normal or inactive mucosal disease is defined as an endoscopy score of 0. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 or who had a missing endoscopy score at Week 44 were considered not to have endoscopic healing. Endoscopy subscore as assessed during central review of video of endoscopy was used.
Time Frame: Week 44
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Participants | 32 | 41 | 51

60. Secondary Outcome: Maintenance Study: Number of Participants With Clinical Remission at Week 44 and Not Receiving Concomitant Corticosteroids at Week 44 Among Participants Who Received Concomitant Corticosteroids at Maintenance Baseline (Per Global Definition)
Description: Global definition of clinical remission: Mayo score <=2 points, with no individual subscore >1. Mayo score includes 4 subscores (stool frequency, rectal bleeding, endoscopy findings, physician's global assessment), rated 0(normal) to 3(severe). Total score=sum of 4 subscores, range: 0 to 12, where 3 to 5=mild; 6 to 10=moderate; 11 to 12=severe; higher scores=worsening of disease. Participants with prohibited change in UC medication/ostomy/colectomy/used rescue medication after clinical flare/ discontinued study drug due to lack of therapeutic effect/AE of worsening of UC before Week 44 considered not to achieved OM of clinical remission and not receiving concomitant corticosteroids (corticosteroid-free clinical remission). Participants with all 4 Mayo subscores missing at Week 44 considered not in clinical remission. Participants missing value in corticosteroid use had their last value carried forward. Endoscopy subscore assessed during central review of video of endoscopy was used.
Time Frame: Week 44
Population: PEAS consisted of all participants who were in clinical response to IV ustekinumab induction and were randomized at Week 0 of the maintenance study to ustekinumab 90 mg SC q8w, ustekinumab 90 mg SC q12w, or placebo SC with, participants who were receiving concomitant corticosteroids at maintenance baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 91 | 82 | 92
Participants | 17 | 25 | 36

61. Secondary Outcome: Maintenance Study: Number of Participants With Clinical Remission at Week 44 and Not Receiving Concomitant Corticosteroids at Week 44 Among Participants Who Received Concomitant Corticosteroids at Maintenance Baseline (Per US Definition)
Description: US definition of clinical remission: absolute stool number <=3, a Mayo rectal bleeding subscore of 0 (no blood seen), and Mayo endoscopy subscore of 0(normal/ inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]), without PGA. Absolute stool number is average of daily stool number over 3 days. Mayo rectal bleeding and endoscopy findings subscores rated as 0 (normal) to 3 (severe). Participants with prohibited change in UC medication/ ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study agent due to lack of therapeutic effect/ AE of worsening of UC before Week 44 or who were missing all 3 of Mayo components related to this OM (absolute stool number, rectal bleeding, and endoscopy subscore) at Week 44 were considered not in clinical remission. Participants with missing value in corticosteroid use had last value carried forward. Endoscopy subscore assessed during central review of video of endoscopy was used.
Time Frame: Week 44
Population: PEAS consisted of all participants who were in clinical response to IV ustekinumab induction and were randomized at Week 0 of the maintenance study to ustekinumab 90 mg SC q8w, ustekinumab 90 mg SC q12w, or placebo SC, with participants who were receiving concomitant corticosteroids at maintenance baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 91 | 82 | 92
Participants | 18 | 27 | 34

62. Secondary Outcome: MS: Change From Maintenance Baseline in Average Daily P.Eq Corticosteroid Dose Through Week 44 Among Participants Who Received Corticosteroids Other Than Budesonide and Beclomethasone Dipropionate at Maintenance Baseline
Description: The change from maintenance baseline in average daily prednisone-equivalent (P.Eq) corticosteroid dose through Week 44 among the participants receiving concomitant corticosteroids other than budesonide and beclomethasone dipropionate at maintenance baseline was reported. Participants who had prohibited change in UC medication/ ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study agent due to lack of therapeutic effect/ AE of worsening of UC before Week 44 had their Week 0 value of the induction study carried forward from the time of the event onward. Participants who had a missing value in corticosteroid use at a timepoint had their last available value carried forward to that timepoint.
Time Frame: Baseline Through Week 44
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: milligram per day (mg/day)
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 75 | 69 | 82
milligram per day (mg/day)
  Change at Week 4 | -7.4 (5.73) | -7.8 (5.48) | -7.2 (5.42)
  Change at Week 8 | -10.8 (6.77) | -11.7 (8.17) | -12.1 (6.81)
  Change at Week 12 | -10.1 (8.71) | -11.6 (9.16) | -12.6 (7.00)
  Change at Week 16 | -10.1 (7.73) | -12.1 (8.37) | -12.8 (6.98)
  Change at Week 20 | -9.5 (7.85) | -12.0 (8.44) | -12.6 (7.27)
  Change at Week 24 | -8.9 (7.96) | -11.9 (8.62) | -12.5 (7.88)
  Change at Week 28 | -7.8 (8.72) | -11.5 (9.23) | -12.4 (7.56)
  Change at Week 32 | -7.7 (8.18) | -11.4 (8.98) | -12.1 (8.21)
  Change at Week 36 | -7.6 (8.28) | -11.3 (8.80) | -11.7 (8.34)
  Change at Week 40 | -7.2 (8.04) | -11.5 (8.62) | -11.5 (8.37)
  Change at Week 44 | -6.8 (7.98) | -11.0 (8.87) | -11.5 (8.37)

63. Secondary Outcome: Maintenance Study: Number of Participants Not Receiving Concomitant Corticosteroids at Week 44 Among Participants Who Received Concomitant Corticosteroids at Maintenance Baseline
Description: Number of participants not receiving concomitant corticosteroids at Week 44 among participants who received concomitant corticosteroids at maintenance Baseline were reported. Participants who had prohibited change in UC medication/ ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study agent due to lack of therapeutic effect/ AE of worsening of UC before Week 44 considered to be receiving concomitant corticosteroids at Week 44. Participants who had a missing value in corticosteroid use at Week 44 had their last value carried forward.
Time Frame: Week 44
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 91 | 82 | 92
Participants | 43 | 56 | 73

64. Secondary Outcome: Maintenance Study: Number of Participants Who Maintained 20-point Improvement From Induction Baseline in IBDQ up to Week 44 Among Participants With a >20-point Improvement in IBDQ at Maintenance Baseline
Description: IBDQ is 32-item questionnaire for participants with IBD used to evaluate disease-specific health-related quality of life. IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). The 32 items were grouped into 4 domains: bowel function, emotional status, systemic symptoms and social function. The 4 domains were scored as:10 to 70 (bowel symptoms); 5 to 35 (systemic symptoms); 12 to 84 (emotional function); and 5 to 35 (social function). For each domain, higher score indicated better quality of life. Total score is sum of each item score and ranges from 32 to 224 with higher score indicating better quality of life. Participants who had prohibited change in UC medication/ ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study agent due to lack of therapeutic effect/ AE of worsening of UC before Week 44 or who had missing IBDQ score were considered not to have maintained improvement in IBDQ.
Time Frame: Up to Week 44
Population: PEAS consisted of all participants who were in clinical response to IV ustekinumab induction and were randomized at Week 0 of the maintenance study to ustekinumab 90 mg SC q8w, ustekinumab 90 mg SC q12w, or placebo SC, with participants with >20-point Improvement in IBDQ at the maintenance baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 129 | 144 | 143
Participants | 64 | 95 | 102

65. Secondary Outcome: Maintenance Study: Change From Maintenance Baseline in the IBDQ Score at Week 20 and 44
Description: IBDQ is 32-item questionnaire for participants with IBD used to evaluate disease-specific health-related quality of life. IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). The 32 items were grouped into 4 domains: bowel function, emotional status, systemic symptoms and social function. The 4 domains were scored as follows: 10 to 70 (bowel symptoms); 5 to 35 (systemic symptoms); 12 to 84 (emotional function); and 5 to 35 (social function). For each domain, higher score indicated better quality of life. Total score is sum of each item score and ranges from 32 to 224 with higher score indicating better quality of life. Participants who had prohibited change in concomitant UC medication or ostomy or colectomy prior to the Week 44 had their Week 0 value of the induction study carried forward from the time of the event onward and participants who had a missing IBDQ score at a timepoint had their last value carried forward.
Time Frame: Baseline, Week 20, and 44
Population: PEAS consisted of all participants who were in clinical response to IV ustekinumab induction and were randomized at Week 0 of the maintenance study to ustekinumab 90 mg SC q8w, ustekinumab 90 mg SC q12w, or placebo SC. Here, n (number of participants analyzed) signifies participants analyzed for this OM at specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Units on a scale
  Change at Week 20: number analyzed (Participants) | 174 | 172 | 174
  Change at Week 20 | -7.0 (31.37) | 0.8 (29.05) | 5.5 (27.40)
  Change at Week 44: number analyzed (Participants) | 173 | 172 | 174
  Change at Week 44 | -15.1 (35.43) | -3.0 (32.89) | 3.9 (31.54)

66. Secondary Outcome: Maintenance Study: Change From Maintenance Baseline in the IBDQ Dimension Scores at Week 20 and 44
Description: The IBDQ is 32-item questionnaire for participants with IBD used to evaluate disease-specific health-related quality of life. IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). The 32 items were grouped into 4 domains: bowel function, emotional status, systemic symptoms and social function. The 4 domains were scored as: 10 to 70 (bowel symptoms); 5 to 35 (systemic symptoms); 12 to 84 (emotional function); 5 to 35 (social function). For each domain, higher score indicated better quality of life. Total score is sum of each item score and ranges from 32 to 224 with higher score indicating better quality of life. Participants who had prohibited change in concomitant UC medication or ostomy or colectomy prior to Week 44 had their Week 0 value of induction study carried forward from time of event onward and participants who had missing IBDQ dimension score at a timepoint had their last available value carried forward.
Time Frame: Baseline, Week 20, and 44
Population: PEAS included all participants who were in clinical response to IV ustekinumab induction and were randomized at Week 0 of the maintenance study to ustekinumab 90 mg SC q8w, ustekinumab 90 mg SC q12w, or placebo SC. Here, n (number of participants analyzed) signifies participants analyzed for this OM for specified categories at specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Units on a scale
  Bowel:Change at Week 20: number analyzed (Participants) | 174 | 172 | 174
  Bowel:Change at Week 20 | -3.2 (10.88) | -0.5 (9.16) | 1.3 (9.56)
  Bowel:Change at Week 44: number analyzed (Participants) | 173 | 172 | 174
  Bowel:Change at Week 44 | -5.7 (12.34) | -1.6 (10.99) | 0.8 (10.49)
  Emotional: Change at Week 20: number analyzed (Participants) | 174 | 172 | 174
  Emotional: Change at Week 20 | -1.9 (12.16) | 0.9 (11.12) | 2.2 (10.56)
  Emotional: Change at Week 44: number analyzed (Participants) | 173 | 172 | 174
  Emotional: Change at Week 44 | -4.7 (13.84) | -0.5 (12.17) | 1.4 (12.22)
  Systemic: Change at Week 20: number analyzed (Participants) | 174 | 172 | 174
  Systemic: Change at Week 20 | -1.1 (5.54) | 0.0 (5.31) | 0.7 (5.24)
  Systemic: Change at Week 44: number analyzed (Participants) | 173 | 172 | 174
  Systemic: Change at Week 44 | -2.2 (5.52) | -0.5 (5.97) | 0.5 (5.83)
  Social: Change at Week 20: number analyzed (Participants) | 174 | 172 | 174
  Social: Change at Week 20 | -0.7 (5.93) | 0.3 (6.59) | 1.4 (5.44)
  Social: Change at Week 44: number analyzed (Participants) | 173 | 172 | 174
  Social: Change at Week 44 | -2.5 (6.72) | -0.5 (7.10) | 1.1 (6.29)

67. Secondary Outcome: Maintenance Study: Change From Maintenance Baseline in 36-Item Short-Form (SF-36) Physical Component Score (PCS) and Mental Component Score (MCS) at Weeks 20 and 44
Description: SF-36 evaluates 8 individual subscales (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, mental health). Each 8 scales scored from 0 to 100 with higher scores= better health. Based on scale scores, PCS (calculated from subscales physical functioning, role-physical, bodily pain, and general health) and MCS (calculated from subscales vitality, social functioning, role-emotional and mental health) scores were derived. Summary MCS and PCS score is also scaled from 0 to 100 with higher scores= better health. Participants with prohibited change in concomitant UC medication/ ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study agent due to lack of therapeutic effect/ due to AE of worsening of UC before Week 44 had Week 0 value of IS carried forward from time of event onward and participants with missing component summary score at timepoint had last available value carried forward.
Time Frame: Baseline, Weeks 20, and 44
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Units on a scale
  PCS: Change at Week 20: number analyzed (Participants) | 173 | 172 | 175
  PCS: Change at Week 20 | -1.2 (6.20) | -0.2 (6.15) | 0.8 (5.55)
  PCS: Change at Week 44: number analyzed (Participants) | 173 | 172 | 175
  PCS: Change at Week 44 | -1.7 (6.45) | -0.4 (7.14) | 1.3 (5.68)
  MCS: Change at Week 20: number analyzed (Participants) | 173 | 172 | 175
  MCS: Change at Week 20 | -1.1 (8.90) | 1.0 (8.91) | 0.4 (9.10)
  MCS: Change at Week 44: number analyzed (Participants) | 173 | 172 | 175
  MCS: Change at Week 44 | -2.4 (9.89) | 0.3 (8.41) | 0.3 (9.51)

68. Secondary Outcome: Maintenance Study: Change From Maintenance Baseline in Individual Subscales of 36-Item Short-Form (SF-36) at Weeks 20 and 44
Description: SF-36 evaluates 8 individual subscales (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health). Each 8 scales scored from 0 to 100 with higher scores= better health. Participants who had prohibited change in concomitant UC medication/ ostomy/ colectomy/ used rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to AE of worsening of UC prior to Week 44 had Week 0 value of induction study carried forward from time of event onward and participants with missing individual scale score at timepoint had last available value carried forward.
Time Frame: Baseline, Weeks 20, and 44
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Units on a scale
  Physical functioning: Change at Week 20: number analyzed (Participants) | 173 | 172 | 175
  Physical functioning: Change at Week 20 | -0.61 (6.140) | -0.01 (5.506) | 0.51 (4.809)
  Physical functioning: Change at Week 44: number analyzed (Participants) | 173 | 172 | 175
  Physical functioning: Change at Week 44 | -1.40 (5.932) | -0.44 (5.624) | 0.66 (4.819)
  Role-physical: Change at Week 20: number analyzed (Participants) | 173 | 172 | 175
  Role-physical: Change at Week 20 | -0.61 (8.630) | 0.17 (7.996) | 0.23 (8.144)
  Role-physical: Change at Week 44: number analyzed (Participants) | 173 | 172 | 175
  Role-physical: Change at Week 44 | -2.27 (9.400) | -0.84 (8.293) | 1.08 (8.096)
  Bodily pain:Change at Week 20: number analyzed (Participants) | 173 | 172 | 175
  Bodily pain:Change at Week 20 | -2.80 (9.081) | -0.30 (8.556) | 1.06 (8.971)
  Bodily pain:Change at Week 44: number analyzed (Participants) | 173 | 172 | 175
  Bodily pain:Change at Week 44 | -2.33 (9.245) | 0.23 (9.340) | 0.94 (8.350)
  General health:Change at Week 20: number analyzed (Participants) | 173 | 172 | 175
  General health:Change at Week 20 | -0.95 (7.468) | 0.67 (7.802) | 1.14 (7.133)
  General health:Change at Week 44: number analyzed (Participants) | 173 | 172 | 175
  General health:Change at Week 44 | -1.62 (7.449) | 0.24 (8.722) | 1.92 (7.955)
  Vitality:Change at Week 20: number analyzed (Participants) | 173 | 172 | 175
  Vitality:Change at Week 20 | -1.71 (8.876) | 0.74 (8.917) | 0.39 (9.209)
  Vitality:Change at Week 44: number analyzed (Participants) | 173 | 172 | 175
  Vitality:Change at Week 44 | -3.18 (10.389) | 0.11 (9.152) | 0.53 (9.743)
  Social functioning: Change at Week 20: number analyzed (Participants) | 173 | 172 | 175
  Social functioning: Change at Week 20 | -0.87 (9.245) | 0.47 (8.979) | 0.72 (9.907)
  Social functioning: Change at Week 44: number analyzed (Participants) | 173 | 172 | 175
  Social functioning: Change at Week 44 | -1.83 (10.186) | 0.06 (9.515) | 1.12 (9.678)
  Role-emotional: Change at Week 20: number analyzed (Participants) | 173 | 172 | 175
  Role-emotional: Change at Week 20 | -0.93 (9.586) | 0.47 (9.338) | 0.14 (8.637)
  Role-emotional: Change at Week 44: number analyzed (Participants) | 173 | 172 | 175
  Role-emotional: Change at Week 44 | -2.21 (10.187) | 0.04 (9.324) | 0.10 (8.199)
  Mental health:Change at Week 20: number analyzed (Participants) | 173 | 172 | 175
  Mental health:Change at Week 20 | -1.07 (9.085) | 1.08 (8.631) | 0.61 (8.467)
  Mental health:Change at Week 44: number analyzed (Participants) | 173 | 172 | 175
  Mental health:Change at Week 44 | -2.15 (9.992) | 0.06 (8.042) | 0.53 (8.915)

69. Secondary Outcome: Maintenance Study: Change From Maintenance Baseline in EuroQOL-5 Dimensions (EQ-5D) Health Questionnaire Index Score at Weeks 20 and 44
Description: EQ-5D descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). The responses to 5 EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 (death) to 1 (full health). Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 had their Week 0 value of the induction study carried forward from the time of the event onward and participants who had a missing individual scale score at a timepoint had their last available value carried forward.
Time Frame: Baseline, Weeks 20, and 44
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Units on a scale
  Change at Week 20: number analyzed (Participants) | 173 | 172 | 175
  Change at Week 20 | -0.036 (0.1535) | -0.002 (0.1694) | 0.016 (0.1471)
  Change at Week 44: number analyzed (Participants) | 173 | 172 | 175
  Change at Week 44 | -0.048 (0.1587) | 0.008 (0.1656) | 0.025 (0.1674)

70. Secondary Outcome: Maintenance Study: Change From Maintenance Baseline in EuroQOL-5 (EQ-5D) Health State Visual Analog Scale (VAS) Score at Weeks 20 and 44
Description: The EQ-5D VAS records the participant's self-rated health on a vertical, VAS, with 0 representing the worst imaginable health state and 100 representing the best imaginable health state. The EQ VAS is used as a quantitative measure of health outcome as judged by the individual participant. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 had their Week 0 value of the induction study carried forward from the time of the event onward and participants who had a missing VAS score at a timepoint had their last available value carried forward.
Time Frame: Baseline, Weeks 20 and 44
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Units on a scale
  Change at Week 20: number analyzed (Participants) | 173 | 172 | 175
  Change at Week 20 | -4.0 (16.70) | -0.3 (17.29) | 2.6 (17.80)
  Change at Week 44: number analyzed (Participants) | 173 | 172 | 175
  Change at Week 44 | -7.7 (18.75) | -2.2 (19.87) | 2.4 (17.28)

71. Secondary Outcome: Maintenance Study: Percentage of Participants With Change From Maintenance Baseline in EuroQOL-5 (EQ-5D) Dimensions Score at Weeks 20 and 44
Description: EQ-5D descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). The responses to 5 EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 (death) to 1 (full health). Participants who had prohibited change in concomitant UC medication/ostomy/ colectomy/ used rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to AE of worsening of UC prior to Week 44 had their Week 0 value of induction study carried forward from time of event onward and who had missing individual scale score at timepoint had their last available value carried forward. Percentage of participants with various responses to the 5 dimensions were reported.
Time Frame: Baseline, Weeks 20, and 44
Population: PEAS consisted of all participants who were in clinical response to IV ustekinumab induction and were randomized at Week 0 of the maintenance study to ustekinumab 90 mg SC q8w, ustekinumab 90 mg SC q12w, or placebo SC. Here, n (number of participants analyzed) signifies participants who were analyzed for this OM at specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
Percentage of participants
  Change at Week (W) 20: Mobility:Improved: number analyzed (Participants) | 173 | 172 | 175
  Change at Week (W) 20: Mobility:Improved | 12.7 | 10.5 | 13.7
  Change at W 20:Mobility:No change: number analyzed (Participants) | 173 | 172 | 175
  Change at W 20:Mobility:No change | 75.7 | 79.1 | 78.9
  Change at W 20:Mobility:Worsened: number analyzed (Participants) | 173 | 172 | 175
  Change at W 20:Mobility:Worsened | 11.6 | 10.5 | 7.4
  Change at W 44:Mobility:Improved: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44:Mobility:Improved | 9.8 | 11.6 | 12.0
  Change at W 44:Mobility:No change: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44:Mobility:No change | 75.1 | 76.2 | 79.4
  Change at W 44:Mobility:Worsened: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44:Mobility:Worsened | 15.0 | 12.2 | 8.6
  Change at W 20:Self-care:Improved: number analyzed (Participants) | 173 | 172 | 174
  Change at W 20:Self-care:Improved | 1.7 | 1.7 | 4.0
  Change at W 20:Self-care:No change: number analyzed (Participants) | 173 | 172 | 174
  Change at W 20:Self-care:No change | 91.9 | 93.6 | 93.7
  Change at W 20:Self-care:Worsened: number analyzed (Participants) | 173 | 172 | 174
  Change at W 20:Self-care:Worsened | 6.4 | 4.7 | 2.3
  Change at W 44:Self-care:Improved: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44:Self-care:Improved | 1.7 | 2.3 | 4.0
  Change at W 44:Self-care:No change: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44:Self-care:No change | 95.4 | 93.0 | 93.1
  Change at W 44:Self-care:Worsened: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44:Self-care:Worsened | 2.9 | 4.7 | 2.9
  Change at W 20:Usual activities:Improved: number analyzed (Participants) | 173 | 172 | 175
  Change at W 20:Usual activities:Improved | 12.7 | 17.4 | 22.3
  Change at W 20:Usual activities:No Change: number analyzed (Participants) | 173 | 172 | 175
  Change at W 20:Usual activities:No Change | 64.2 | 66.9 | 64.0
  Change at W 20:Usual activities:Worsened: number analyzed (Participants) | 173 | 172 | 175
  Change at W 20:Usual activities:Worsened | 23.1 | 15.7 | 13.7
  Change at W 44: Usual activities:Improved: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44: Usual activities:Improved | 14.5 | 24.4 | 25.1
  Change at W 44:Usual activities:No Change: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44:Usual activities:No Change | 52.6 | 55.2 | 62.9
  Change at W 44:Usual activities:Worsened: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44:Usual activities:Worsened | 32.9 | 20.3 | 12.0
  Change at W 20:Pain/discomfort: Improved: number analyzed (Participants) | 173 | 172 | 175
  Change at W 20:Pain/discomfort: Improved | 16.8 | 22.1 | 23.4
  Change at W 20:Pain/discomfort: No Change: number analyzed (Participants) | 173 | 172 | 175
  Change at W 20:Pain/discomfort: No Change | 54.9 | 58.7 | 58.9
  Change at W 20:Pain/discomfort: Worsened: number analyzed (Participants) | 173 | 172 | 175
  Change at W 20:Pain/discomfort: Worsened | 28.3 | 19.2 | 17.7
  Change at W 44:Pain/discomfort: Improved: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44:Pain/discomfort: Improved | 17.9 | 25.0 | 30.3
  Change at W 44:Pain/discomfort: No Change: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44:Pain/discomfort: No Change | 46.2 | 55.8 | 50.9
  Change at W 44:Pain/discomfort: Worsened: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44:Pain/discomfort: Worsened | 35.8 | 19.2 | 18.9
  Change at W 20:Anxiety/depression: Improved: number analyzed (Participants) | 173 | 172 | 175
  Change at W 20:Anxiety/depression: Improved | 16.2 | 20.3 | 24.6
  Change at W 20:Anxiety/depression: No Change: number analyzed (Participants) | 173 | 172 | 175
  Change at W 20:Anxiety/depression: No Change | 62.4 | 61.6 | 58.3
  Change at W 20:Anxiety/depression: Worsened: number analyzed (Participants) | 173 | 172 | 175
  Change at W 20:Anxiety/depression: Worsened | 21.4 | 18.0 | 17.1
  Change at W 44:Anxiety/depression: Improved: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44:Anxiety/depression: Improved | 17.9 | 20.3 | 26.9
  Change at W 44:Anxiety/depression: No Change: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44:Anxiety/depression: No Change | 56.1 | 58.7 | 58.9
  Change at W 44:Anxiety/depression: Worsened: number analyzed (Participants) | 173 | 172 | 175
  Change at W 44:Anxiety/depression: Worsened | 26.0 | 20.9 | 14.3

72. Secondary Outcome: Maintenance Study: Number of Participants With Mucosal Healing at Week 44
Description: Mucosal healing included EH and HH. EH: endoscopy subscore of 0 (normal/ inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]). HH: neutrophil infiltration in <5% of crypts, no crypt destruction, no erosions/ ulcerations/ granulation tissue. Participants with prohibited change in concomitant UC medication/ ostomy/ colectomy/ used rescue medication after clinical flare/ discontinued study agent due to lack of therapeutic effect/ due to AE of worsening of UC prior to Week 44/ missing endoscopy score/ missing any component of histologic healing (i.e. assessment of neutrophils in crypts, crypt destruction/ erosions/ ulcerations/ granulations) at Week 44 and had unevaluable biopsy (biopsy collected but could not assessed due to sample preparation/ technical errors) at Week 44, but who did not achieve endoscopic healing, considered not to have mucosal healing. Endoscopy subscore assessed during central review used endoscopy video.
Time Frame: Week 44
Population: PEAS consisted of all participants who were in clinical response to IV ustekinumab induction and were randomized at Week 0 of the maintenance study to ustekinumab 90 mg SC q8w, ustekinumab 90 mg SC q12w, or placebo SC, with participants whose mucosal healing status was determined at Week 44 with evaluable biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 170 | 170 | 172
Participants | 41 | 66 | 79

73. Secondary Outcome: Maintenance Study: Change From Maintenance Baseline in C-reactive Protein (CRP) Concentration at Weeks 8, 24, and 44
Description: Change from Maintenance baseline in CRP concentration at Weeks 8, 24, and 44 were reported. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 had their Week 0 value of the induction study carried forward from the time of the event onward. Participants who had a missing CRP value at the designated analysis timepoint had their last value carried forward.
Time Frame: Baseline, Weeks 8, 24, and 44
Population: as for outcome 71
Measure: Median (Inter-Quartile Range); unit: milligram per liter (mg/L)
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
milligram per liter (mg/L)
  Change at Week 8: number analyzed (Participants) | 174 | 170 | 176
  Change at Week 8 | 0.05 [-0.67 to 0.81] | -0.03 [-0.92 to 0.37] | -0.04 [-1.50 to 0.92]
  Change at Week 24: number analyzed (Participants) | 174 | 170 | 176
  Change at Week 24 | 0.68 [-0.28 to 2.34] | 0.13 [-0.75 to 1.16] | -0.03 [-1.53 to 0.59]
  Change at Week 44: number analyzed (Participants) | 174 | 170 | 175
  Change at Week 44 | 1.07 [0.00 to 5.18] | 0.38 [-0.35 to 1.53] | -0.07 [-1.73 to 0.79]

74. Secondary Outcome: Maintenance Study: Change From Maintenance Baseline in Fecal Lactoferrin Concentration at Weeks 8, 24, and 44
Description: Change from Maintenance baseline in fecal lactoferrin concentration at Weeks 8, 24, and 44 were reported. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 had their Week 0 value of the induction study carried forward from the time of the event onward. Participants who had a missing fecal lactoferrin value at the designated analysis timepoint had their last value carried forward.
Time Frame: Baseline, Weeks 8, 24, and 44
Population: as for outcome 71
Measure: Median (Inter-Quartile Range); unit: microgram per gram (mcg/g)
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
microgram per gram (mcg/g)
  Change at Week 8: number analyzed (Participants) | 167 | 161 | 163
  Change at Week 8 | 0.0 [-44.8 to 72.0] | 0.0 [-35.0 to 48.5] | -1.4 [-52.0 to 30.9]
  Change at Week 24: number analyzed (Participants) | 166 | 161 | 161
  Change at Week 24 | 2.2 [-45.3 to 139.9] | -0.8 [-47.9 to 35.1] | -2.3 [-65.5 to 25.5]
  Change at Week 44: number analyzed (Participants) | 166 | 159 | 160
  Change at Week 44 | 0.8 [-34.2 to 177.4] | -1.9 [-54.4 to 35.1] | -9.1 [-101.6 to 7.8]

75. Secondary Outcome: Maintenance Study: Change From Maintenance Baseline in Fecal Calprotectin Concentration at Weeks 8, 24, and 44
Description: Change from Maintenance baseline in fecal calprotectin concentration at Weeks 8, 24, and 44 were reported. Participants who had a prohibited change in concomitant UC medication or an ostomy or colectomy, or used a rescue medication after clinical flare, or discontinued study agent due to lack of therapeutic effect or due to an AE of worsening of UC prior to the Week 44 had their Week 0 value of the induction study carried forward from the time of the event onward. Participants who had a missing fecal calprotectin value at the designated analysis timepoint had their last value carried forward.
Time Frame: Baseline, Weeks 8, 24, and 44
Population: as for outcome 71
Measure: Mean (Inter-Quartile Range); unit: milligram per kilogram (mg/kg)
Arm/Group | Maintenance Study (MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90 mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90 mg SC Every 8 Weeks (q8w)
Number analyzed (Participants) | 175 | 172 | 176
milligram per kilogram (mg/kg)
  Change at Week 8: number analyzed (Participants) | 168 | 160 | 161
  Change at Week 8 | 0.0 [-158.0 to 557.0] | -18.5 [-368.5 to 225.5] | -31.0 [-380.0 to 205.0]
  Change at Week 24: number analyzed (Participants) | 165 | 160 | 159
  Change at Week 24 | 125.0 [-97.0 to 1223.0] | -31.5 [-413.5 to 385.0] | -46.0 [-530.0 to 318.0]
  Change at Week 44: number analyzed (Participants) | 164 | 158 | 159
  Change at Week 44 | 229.5 [-102.5 to 1387.0] | -37.5 [-476.0 to 274.0] | -85.0 [-742.0 to 166.0]

ADVERSE EVENTS:
Time Frame: Up to Week 220
Description: The safety analysis set included participants who received at least 1 dose of study agent, including partial dose, according to actual treatment received.
Groups:
- IS: Placebo-Nonresponders at Week 8: Participants who did not achieve clinical response to placebo IV at Week 8 and received a single IV infusion of ustekinumab approximating 6 mg/kg at Week 8. Included data from Week 8 onward through the final safety visit.
- IS: Ustekinumab Nonresponders at Week 8: Participants who did not achieve clinical response to ustekinumab (130 mg or approximately 6 mg/kg [IV]) at Week 8 and received a single dose of ustekinumab 90 mg SC along with matching placebo IV (to maintain the blind). Participants with clinical response at Week 16 (that is, delayed responders) were eligible to enter Maintenance study, but were not be randomized. Included data from Week 8 onward through the final safety visit.
- LTE: Placebo SC to Ustekinumab SC 90 mg q8w: Participants who were randomized to receive placebo SC in the maintenance study and had a dose adjustment from placebo SC to ustekinumab 90 mg SC every 8 weeks (q8w) during the LTE.
- LTE: Ustekinumab 90 mg SC q12w to 90 mg SC q8w: Participants who received ustekinumab 90 mg SC every 12 weeks (q12w) completed the maintenance Week 44 visit and benefited from continued treatment entered the LTE period, and received ustekinumab 90 mg at Week 48 until Week 220.
- LTE: Ustekinumab 90 mg SC q8w to 90 mg SC q8w: Participants who were randomized to receive ustekinumab 90 mg SC q8w in the maintenance study and had a sham dose adjustment to ustekinumab 90 mg SC q8w during the LTE.
Arm/Group | Induction Study(IS): Placebo Intravenous (IV) | IS: Ustekinumab 130 Milligram (mg) IV | IS: Ustekinumab Approximately 6mg/kg IV | IS: Placebo-Nonresponders at Week 8 | IS: Ustekinumab Nonresponders at Week 8 | Maintenance Study(MS): Placebo Subcutaneous (SC) | MS: Ustekinumab 90mg SC Every 12 Weeks (q12w) | MS: Ustekinumab 90mg SC Every 8 Weeks (q8w) | MS: Placebo IV (IS - Responders) to Placebo SC | MS: Ustekinumab Delayed Responders(IS) to UST 90mg SC q8w | Long Term Extension (LTE): Placebo SC | LTE: Placebo SC to Ustekinumab SC 90 mg q8w | LTE: Ustekinumab 90 mg SC q12w | LTE: Ustekinumab 90 mg SC q12w to 90 mg SC q8w | LTE: Ustekinumab 90 mg SC q8w | LTE: Ustekinumab 90 mg SC q8w to 90 mg SC q8w | LTE: Placebo IV (IS - Responders) to Placebo SC | LTE: Ustekinumab Delayed Responders (IS) to UST 90mg SC q8w
All-Cause Mortality (participants affected / at risk) | 0/319 | 0/321 | 1/320 | 0/184 | 0/233 | 0/175 | 0/172 | 0/176 | 0/103 | 1/157 | 0/115 | 1/56 | 0/141 | 0/64 | 0/143 | 0/37 | 0/73 | 0/116
Serious Adverse Events (participants affected / at risk) | 22/319 | 12/321 | 11/320 | 7/184 | 12/233 | 17/175 | 13/172 | 15/176 | 8/103 | 11/157 | 6/115 | 8/56 | 13/141 | 6/64 | 15/143 | 3/37 | 10/73 | 14/116
Other Adverse Events (participants affected / at risk) | 91/319 | 100/321 | 103/320 | 27/184 | 30/233 | 121/175 | 93/172 | 118/176 | 69/103 | 93/157 | 68/115 | 48/56 | 98/141 | 38/64 | 105/143 | 27/37 | 45/73 | 91/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Study(IS): Placebo Intravenous (IV) (N=319) | IS: Ustekinumab 130 Milligram (mg) IV (N=321) | IS: Ustekinumab Approximately 6mg/kg IV (N=320) | IS: Placebo-Nonresponders at Week 8 (N=184) | IS: Ustekinumab Nonresponders at Week 8 (N=233) | Maintenance Study(MS): Placebo Subcutaneous (SC) (N=175) | MS: Ustekinumab 90mg SC Every 12 Weeks (q12w) (N=172) | MS: Ustekinumab 90mg SC Every 8 Weeks (q8w) (N=176) | MS: Placebo IV (IS - Responders) to Placebo SC (N=103) | MS: Ustekinumab Delayed Responders(IS) to UST 90mg SC q8w (N=157) | Long Term Extension (LTE): Placebo SC (N=115) | LTE: Placebo SC to Ustekinumab SC 90 mg q8w (N=56) | LTE: Ustekinumab 90 mg SC q12w (N=141) | LTE: Ustekinumab 90 mg SC q12w to 90 mg SC q8w (N=64) | LTE: Ustekinumab 90 mg SC q8w (N=143) | LTE: Ustekinumab 90 mg SC q8w to 90 mg SC q8w (N=37) | LTE: Placebo IV (IS - Responders) to Placebo SC (N=73) | LTE: Ustekinumab Delayed Responders (IS) to UST 90mg SC q8w (N=116)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Autoimmune Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deafness Neurosensory (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness Unilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal Detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal Fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorectal Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 11 | 4 | 4 | 5 | 4 | 8 | 1 | 2 | 3 | 7 | 3 | 2 | 1 | 3 | 5 | 1 | 4 | 2
Colon Dysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterovesical Fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mesenteric Fibrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pseudopolyposis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver Disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Clostridium Difficile Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Complicated Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus Colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis Salmonella (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Human Herpesvirus 6 Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Listeriosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic Inflammatory Disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Periorbital Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perirectal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngeal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pneumonia Legionella (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salpingitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salpingo-Oophoritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bladder Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaw Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural Intestinal Perforation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intraductal Papilloma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lentigo Maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testis Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Motor Dysfunction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Optic Neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Calculus Bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glomerulonephritis Chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary Eosinophilia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyoderma Gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extremity Necrosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Study(IS): Placebo Intravenous (IV) (N=319) | IS: Ustekinumab 130 Milligram (mg) IV (N=321) | IS: Ustekinumab Approximately 6mg/kg IV (N=320) | IS: Placebo-Nonresponders at Week 8 (N=184) | IS: Ustekinumab Nonresponders at Week 8 (N=233) | Maintenance Study(MS): Placebo Subcutaneous (SC) (N=175) | MS: Ustekinumab 90mg SC Every 12 Weeks (q12w) (N=172) | MS: Ustekinumab 90mg SC Every 8 Weeks (q8w) (N=176) | MS: Placebo IV (IS - Responders) to Placebo SC (N=103) | MS: Ustekinumab Delayed Responders(IS) to UST 90mg SC q8w (N=157) | Long Term Extension (LTE): Placebo SC (N=115) | LTE: Placebo SC to Ustekinumab SC 90 mg q8w (N=56) | LTE: Ustekinumab 90 mg SC q12w (N=141) | LTE: Ustekinumab 90 mg SC q12w to 90 mg SC q8w (N=64) | LTE: Ustekinumab 90 mg SC q8w (N=143) | LTE: Ustekinumab 90 mg SC q8w to 90 mg SC q8w (N=37) | LTE: Placebo IV (IS - Responders) to Placebo SC (N=73) | LTE: Ustekinumab Delayed Responders (IS) to UST 90mg SC q8w (N=116)
Anaemia (Blood and lymphatic system disorders) | 11 | 7 | 8 | 4 | 1 | 12 | 7 | 7 | 9 | 9 | 1 | 3 | 4 | 3 | 2 | 1 | 3 | 4
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 5 | 0 | 1 | 3 | 2 | 3 | 4 | 5 | 0 | 2 | 3 | 0 | 0 | 0 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 3 | 4 | 1 | 2 | 1 | 0 | 2 | 0 | 0 | 3
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 3 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 4 | 2 | 5 | 1 | 1 | 0 | 3 | 2 | 0 | 5 | 0 | 0 | 3
Abdominal Pain (Gastrointestinal disorders) | 9 | 8 | 5 | 0 | 0 | 4 | 6 | 8 | 3 | 5 | 2 | 1 | 2 | 2 | 15 | 1 | 4 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 4 | 1 | 0 | 2 | 1 | 0 | 4 | 1 | 1 | 3 | 2 | 4 | 1 | 2 | 1 | 1 | 2
Colitis Ulcerative (Gastrointestinal disorders) | 8 | 5 | 5 | 1 | 3 | 48 | 19 | 16 | 25 | 23 | 23 | 11 | 34 | 20 | 37 | 13 | 27 | 30
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 6 | 0 | 3 | 1 | 0 | 1 | 1 | 1 | 0 | 5 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 0 | 2 | 5 | 7 | 2 | 6 | 2 | 1 | 6 | 3 | 13 | 2 | 4 | 9
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 7 | 8 | 7 | 3 | 3 | 4 | 4 | 6 | 3 | 5 | 2 | 1 | 5 | 1 | 9 | 1 | 1 | 5
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 4 | 0 | 3 | 5 | 1 | 1 | 0 | 3 | 3 | 2 | 0 | 1 | 6 | 0 | 0 | 2
Fatigue (General disorders) | 5 | 6 | 8 | 0 | 1 | 4 | 4 | 7 | 3 | 3 | 4 | 1 | 0 | 2 | 5 | 1 | 1 | 2
Influenza Like Illness (General disorders) | 2 | 2 | 1 | 1 | 1 | 4 | 2 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 4 | 0 | 1 | 5
Injection Site Erythema (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 3 | 0 | 0 | 1 | 0 | 5 | 1 | 0 | 3
Injection Site Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Pyrexia (General disorders) | 6 | 4 | 6 | 1 | 0 | 7 | 1 | 8 | 5 | 5 | 2 | 3 | 0 | 0 | 1 | 0 | 2 | 7
Hepatic Steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 1 | 0 | 6 | 5 | 6 | 5 | 6 | 2 | 3 | 7 | 2 | 4 | 0 | 0 | 6
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 4
Ear Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 5 | 5 | 7 | 2 | 5 | 1 | 2 | 4 | 0 | 5 | 3 | 2 | 8
Herpes Zoster (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 5
Influenza (Infections and infestations) | 0 | 2 | 1 | 0 | 2 | 8 | 5 | 10 | 6 | 7 | 4 | 4 | 6 | 3 | 10 | 3 | 6 | 3
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 9 | 13 | 18 | 7 | 1 | 28 | 31 | 26 | 13 | 19 | 17 | 13 | 29 | 10 | 27 | 12 | 5 | 32
Oral Herpes (Infections and infestations) | 5 | 1 | 3 | 0 | 0 | 1 | 1 | 3 | 2 | 0 | 0 | 1 | 3 | 1 | 6 | 2 | 4 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 2 | 3 | 2 | 4 | 2 | 1 | 0 | 3 | 1 | 3 | 2 | 3 | 0
Rhinitis (Infections and infestations) | 0 | 3 | 1 | 1 | 1 | 2 | 2 | 4 | 0 | 1 | 2 | 2 | 2 | 1 | 2 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 5 | 1 | 0 | 1 | 2 | 2 | 7 | 1 | 3 | 3 | 2 | 5 | 1 | 8 | 4 | 1 | 4
Tonsillitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 2 | 0 | 1 | 1 | 3 | 0 | 3 | 1 | 1 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 6 | 5 | 2 | 5 | 8 | 5 | 16 | 4 | 7 | 6 | 4 | 12 | 4 | 17 | 2 | 4 | 10
Urinary Tract Infection (Infections and infestations) | 0 | 3 | 3 | 1 | 0 | 4 | 3 | 2 | 2 | 4 | 2 | 2 | 0 | 3 | 6 | 3 | 1 | 3
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 3 | 1 | 1 | 2 | 0 | 3 | 0 | 3 | 2 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 4 | 0 | 1 | 0 | 2 | 1 | 0 | 3 | 0 | 0 | 2
Heat Illness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 2
Alanine Aminotransferase Increased (Investigations) | 2 | 0 | 6 | 0 | 0 | 4 | 5 | 6 | 3 | 1 | 0 | 7 | 3 | 3 | 3 | 1 | 0 | 4
Aspartate Aminotransferase Increased (Investigations) | 2 | 0 | 3 | 0 | 0 | 4 | 5 | 4 | 4 | 3 | 0 | 5 | 1 | 3 | 4 | 1 | 0 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Blood Phosphorus Decreased (Investigations) | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Stool Analysis Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 3 | 2 | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 4 | 2 | 0 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 5 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 6 | 1 | 2 | 17 | 16 | 10 | 9 | 16 | 6 | 4 | 9 | 5 | 11 | 2 | 4 | 10
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 4 | 0 | 1 | 7 | 1 | 7 | 3 | 5 | 5 | 6 | 7 | 3 | 7 | 2 | 5 | 6
Dizziness (Nervous system disorders) | 1 | 2 | 4 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 14 | 22 | 13 | 2 | 2 | 7 | 11 | 18 | 4 | 9 | 7 | 4 | 9 | 2 | 11 | 2 | 4 | 11
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 2
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 1 | 0 | 1 | 0 | 2 | 3 | 3 | 4 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3 | 0 | 0 | 5 | 2 | 7 | 4 | 4 | 5 | 5 | 2 | 2 | 7 | 1 | 1 | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 8 | 1 | 0 | 5 | 4 | 7 | 1 | 1 | 0 | 1 | 7 | 0 | 5 | 0 | 1 | 3
Acne (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 0 | 0 | 0 | 2 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 5 | 1 | 2 | 0 | 1 | 5 | 0 | 3 | 2 | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 0 | 3
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 8 | 3 | 1 | 0 | 4 | 1 | 2 | 3 | 2 | 1 | 1 | 1 | 2 | 2 | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 4 | 1 | 2 | 6 | 6 | 6 | 2 | 2 | 0 | 1 | 2 | 1 | 5 | 1 | 6 | 3
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 5 | 1 | 0 | 0 | 0 | 0 | 4 | 3 | 1 | 3 | 1 | 2 | 5 | 1 | 5 | 3 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT02407236/Prot_002.pdf
  • Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT02407236/SAP_001.pdf